| | Statistical Analysis Plan Final |
|---|---|
| <b>gsk</b> GlaxoSmithKline | Statistical Analysis Plan |
| Detailed Title: | A Phase 1/2 randomised observer-blind placebo-<br>controlled study to evaluate the safety, reactogenicity<br>and immunogenicity of different dose levels of GSK<br>Biologicals' investigational unadjuvanted RSV<br>maternal vaccine (GSK3888550A) compared to<br>placebo when administered to healthy non-pregnant<br>women aged 18-45 years |
| eTrack study number and<br>Abbreviated Title | 208068 (RSV-MAT-001) |
| Scope: | All data pertaining to the above study |
| Date of Statistical Analysis<br>Plan | Final: 25-Oct-2018 |
| Co-ordinating author: | (Expert Biostatistician) |
| Reviewed by: | PPD (Clinical and Epidemiology Project Lead) PPD (Clinical Research and Development Lead) PPD (Lead statistician) PPD (Lead statistical analyst) PPD (Scientific writer) PPD (Regulatory Affair) PPD (SERM physician) PPD (Public disclosure representative) |
| Approved by: | (Clinical and Epidemiology Project Lead); PPD (Clinical Research and Development Lead); PPD (Lead statistician); PPD (Lead stat Analyst); PPD (Study Statistician) |

APP 9000058193 Statistical Analysis Plan Template (Effective date: 14 April 2017)

208068 (RSV-MAT-001) Statistical Analysis Plan Final

# **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| LIS | ST OF A | BBREVIATIONS. | | 11 |
| 1. | DOC | JMENT HISTORY | | 12 |
| 2. | STUE | Y DESIGN | | 12 |
| 3. | OD IE | CTIVES | | 1.1 |
| ა. | 3.1. | | ) | |
| | 3.1. | | tive | |
| | 3.3. | | ÷ | |
| 4. | ENDE | POINTS | | 1/ |
| →. | 4.1. | | ts | |
| | 4.2. | | oints | |
| | 4.3. | | | |
| | | , , | | |
| 5. | | | | |
| | 5.1. | | | |
| | | | ed Set (ES) | |
| | | | otocol set (PPS) for analysis of immunogenicity | |
| | 5.2. | | nating data from Analysis Sets | |
| | | | tion from Exposed Set (ES) | |
| | | | tion from Per-protocol analysis Set (PPS) | |
| | | 5.2.2.1 | . Excluded subjects | 17 |
| | | 5.2.2.2 | . Right censored Data | 17 |
| | | | . Visit-specific censored Data | 18 |
| | 5.3. | Important protoco protocol analysis | ol deviation not leading to elimination from per-<br>set | 19 |
| _ | 0.7.4.7 | IOTIONI ANIALYO | | 4.0 |
| 6. | | | ES | |
| | 6.1. | Demography 6.1.1. Analysi | s of demographics/baseline characteristics planned | 19 |
| | | | rotocol | 10 |
| | | | nal considerations | |
| | 6.2. | | ilai considerations | |
| | 0.2. | | is of exposure planned in the protocol | |
| | 6.3. | • | s of exposure planned in the protocor | |
| | 0.5. | | s of immunogenicity planned in the protocol | |
| | | 6.3.1.1 | | |
| | | 6.3.1.2 | | |
| | | | nal considerations | |
| | 6.4. | | y | |
| | U. <del>4</del> . | | is of safety planned in the protocol | |
| | | 6.4.1.1 | • | |
| | | | nal considerations | |
| | | 6.4.2.1 | | 20 |
| | | 0.7.2.1 | Event | 26 |
| | | 6.4.2.2 | | 20 |
| | | U. 1.Z.Z | Events | 26 |
| | | | — : -:- <del></del> | |

| | Statistical Arialy | SIS FIAITI IIIAI |
|---|---|---|
| 7. | ANALYSIS INTERPRETATION | <mark>26</mark> |
| 8. | CONDUCT OF ANALYSES | 27 |
| | 8.1. Sequence of analyses | <mark>27</mark> |
| | 8.2. Statistical considerations for interim analyses | |
| 9. | CHANGES FROM PLANNED ANALYSES | 28 |
| 10. | LIST OF FINAL REPORT TABLES, LISTINGS AND FIGURES | 28 |
| 11. | ANNEX 1 STANDARD DATA DERIVATION RULE AND STATISTICAL | 20 |
| | METHODS | |
| | 11.1. Statistical Method References | |
| | 11.2. Standard data derivation | |
| | 11.2.1. Date derivation | |
| | 11.2.2. Demography | |
| | 11.2.3. Immunogenicity | |
| | 11.2.4. Safety | 31 |
| | 11.2.5. Number of decimals displayed: | 32 |
| 12. | ANNEX 2: TOXICITYGRADING SCALE FOR LABORATORY | |
| | ASSESSMENTS | 32 |
| 13. | ANNEX 3: STUDY SPECIFIC MOCK TFL | 33 |
| | 13.1. List of individual data listing | |
| | 13.2. Template of Tables and Figures | |

208068 (RSV-MAT-001) Statistical Analysis Plan Final

# **LIST OF TABLES**

| | | PAGE |
|---------|---------------------------------------------------------|------|
| Table 1 | Blinding of study epochs | 13 |
| Table 2 | Intervals between study visits | 16 |
| Table 3 | Implausible Solicited Adverse Events | 26 |
| Table 4 | FDA toxicity grading scales for biochemistry parameters | 32 |
| Table 5 | FDA toxicity grading scales for hematology parameters | 33 |

208068 (RSV-MAT-001) Statistical Analysis Plan Final

# **LIST OF FIGURES**

| | | PAGE |
|----------|--------------|------|
| Figure 1 | Study Design | 12 |

208068 (RSV-MAT-001) Statistical Analysis Plan Final

# **LIST OF TEMPLATES**

| | | PAGE |
|---|---|---|
| Template 1 | Number of subjects by country and center <exposed set=""></exposed> | 35 |
| Template 2 | Number of subjects vaccinated, completed and withdrawn with reason for withdrawal – up to <day 31,="" 91,="" day="" end="" study=""> <exposed set=""></exposed></day> | 35 |
| Template 3 | Visit attendance – up to <day 31,="" 91,="" day="" end="" study=""> <exposed set=""></exposed></day> | 35 |
| Template 4 | Summary of important protocol deviation leading to elimination from Per protocol set <enrolled set=""></enrolled> | 36 |
| Template 5 | Consort flow - Part 1 from enrolment to randomization <all enrolled="" set=""></all> | 36 |
| Template 6 | Consort – Part II from randomization to exposure for each study group <all randomised="" set=""></all> | 37 |
| Template 7 | Consort flow - Part 3 from exposure to per protocol set, per study group <exposed set=""></exposed> | 37 |
| Template 8 | Summary of demographic characteristics <exposed 31,="" 61,="" 91="" <8,="" at="" day="" for="" immunogenicity="" pps="" set,="">&gt;</exposed> | 38 |
| Template 9 | Summary of vital signs characteristics <exposed 31,="" 61,="" 91="" <8,="" at="" day="" for="" immunogenicity="" pps="" set,="">&gt;</exposed> | 39 |
| Template 10 | Deviations from specifications for age and intervals between study visits <exposed set=""></exposed> | 40 |
| Template 11 | Study Population – Up to <day 91,="" end="" study=""> <exposed set=""></exposed></day> | 41 |
| Template 12 | Number of enrolled subjects by country | 41 |
| Template 13 | Number of enrolled subjects by age category | 41 |
| Template 14 | Minimum and maximum activity dates <exposed set=""></exposed> | 42 |
| Template 15 | Compliance in completing solicited symptoms information <exposed set=""></exposed> | 42 |
| Template 16 | Incidence and nature of <any, 2="" 3="" 3,="" and="" grade="" related,=""> adverse events (unsolicited and solicited) <requiring attention="" medical=""> reported during the &lt;7,30&gt;-days (Day 1-&lt;7,30&gt;) post-vaccination period <exposed set=""></exposed></requiring></any,> | 42 |
| Template 17 | Incidence of solicited local adverse events reported during the 7-day (Days 1-7) post-vaccination period by maximum grading <exposed set=""></exposed> | 43 |

| Template 18 | Number of days with solicited local adverse event during the 7-day (Days 1-7) post-vaccination period <exposed set="">4</exposed> |
|---|---|
| Template 19 | Percentage of subjects reporting solicited local adverse events (any grade /grade 2,3/ grade 3) during the 7-day (Days 1-7) post-vaccination period by maximum intensity <exposed set="">48</exposed> |
| Template 20 | Incidence of solicited general adverse event reported during the 7-day (Days 1-7) post-vaccination period by maximum grading <exposed set=""></exposed> |
| Template 21 | Number of days with solicited general adverse event during the 7-day (Days 1-7) post-vaccination period <exposed set="">4</exposed> |
| Template 22 | Percentage of subjects reporting fever (any and grade 3) and other solicited general adverse events (any grade /grade 2,3/ grade 3) during the 7-day (Days 1-7) post-vaccination period by maximum intensity <exposed set=""></exposed> |
| Template 23 | Percentage of subjects reporting the occurrence of <any, 3="" grade=""> <unsolicited adverse="" events="" serious="" symptoms,=""> classified by MedDRA Primary System Organ Class and Preferred Term <with attended="" causal="" medically="" relationship="" to="" vaccination,="" visit="" with="">, within the 30-day (Days 1-30) post-vaccination period <exposed set=""></exposed></with></unsolicited></any,> |
| Template 24 | Percentage of subjects reporting the occurrence of <serious adverse="" events=""> classified by MedDRA Primary System Organ Class and Preferred Term from <vaccination 91="" day="" end="" from="" study="" to="" up="" vaccination="" visit,=""> <exposed set=""></exposed></vaccination></serious> |
| Template 25 | Number and percentage of subjects taking a concomitant medication <during <7,30="" the="">- day (Days 1-&lt;7,30&gt;) post-vaccination period, from vaccination to Day 91 visit/study end&gt; <exposed set=""></exposed></during> |
| Template 26 | Distribution of change from baseline in hematology and biochemistry with respect to normal laboratory ranges <exposed set=""></exposed> |
| Template 27 | Summary of hematology and biochemistry results by maximum grade up to <visit (d31)="" (d8),="" 2="" 3="" visit=""> post vaccination versus baseline <exposed set=""></exposed></visit> |
| Template 28 | Summary of haematology change from baseline by maximum grade in the specified category <up (d31)="" (d8),="" 3="" to="" up="" visit="" visit2=""><exposed set=""></exposed></up> |
| Template 29 | Individuals results of <hemoglobin 2,="" <equal="" above="" alt,="" and="" ast,="" blood="" cells,="" count="" count,="" creatinine,="" grade="" higher="" levels,="" ll="" ll,="" lower="" nitrogen="" normal="" outside="" platelet="" range,="" than="" the="" urea="" white="">&lt; group&gt; <exposed set=""></exposed></hemoglobin> |

| Template 30 | Solicited and unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term within the 30- day (Days 1-30) post-vaccination period including number of events - SAE excluded <exposed set=""></exposed> | 53 |
|---|---|---|
| Template 31 | Number (%) of subjects with serious adverse events including number of events reported <within (days="" 1-30)="" 30="" days="" period="" post="" vaccination=""><from 91="" day="" end="" study="" to="" up="" vaccination="" visit,=""> <exposed set=""></exposed></from></within> | 54 |
| Template 32 | Listing of all SAEs <within (days="" 1-30)="" 30="" 91,="" <day="" day="" end="" from="" period,="" post-vaccination="" study="" to="" up="" vaccination=""> &gt;<exposed set=""></exposed></within> | 55 |
| Template 33 | Listing of adverse events, SAEs and solicited symptoms leading to withdrawal from the study <within (days="" 1-30)="" 30="" days="" period="" post-vaccination=""><during 91,="" <day="" end="" study="" to="" up="" vaccination=""> <exposed set=""></exposed></during></within> | 55 |
| Template 34 | Listing of all pregnancies from vaccination up to study end <exposed set=""></exposed> | 56 |
| Template 35 | Number and percentage of subjects with <rsv-a antibody="" concentration="" igg="" neutralising="" rsv="" titre,=""> equal to or above <cut-off> and <gmts gmcs=""> <pps exposed="" for="" immunogenicity,="" set=""></pps></gmts></cut-off></rsv-a> | 57 |
| Template 36 | Distribution of RSV-A neutralising antibody titre <pps <at="" day="" for="" immunogenicity="" x="">&gt;</pps> | 58 |
| Template 37 | Distribution of fold of anti-RSV-A neutralising antibody titre by pre-vaccination titre category <pps for="" immunogenicity=""></pps> | 58 |
| Template 38 | Geometric mean of the individual ratio of <rsv-a antibody="" concentrations="" igg="" neutralizing="" rsv="" titres,=""> at <day 31,="" 61,="" 8,="" 91="" day=""> compared to pre-vaccination with 95% CI <pps 31="" day="" for="" immunogenicity<at="">&gt;</pps></day></rsv-a> | 59 |
| Template 39 | Estimated <gmts,gmcs> and 95% CIs for <rsv-a antibody="" concentration="" igg="" neutralising="" rsv="" titre,=""> (PPS for immunogenicity)</rsv-a></gmts,gmcs> | 60 |
| Template 40 | <gmts, gmcs=""> and their 95% CIs for <rsv-a antibody="" concentration="" igg="" neutralising="" rsv="" titres,=""> at each timepoint up to Day &lt;31,91&gt; <pps for="" immunogenicity=""></pps></rsv-a></gmts,> | 61 |
| Template 41 | Reverse cumulative distribution curves for <anti-rsv-a antibody="" concentrations="" igg="" neutralising="" rsv="" titres,=""> in each group at pre-vaccination and <day 31,="" 61,="" 8,="" 91="" day=""> <pps for="" immunogenicity=""></pps></day></anti-rsv-a> | 62 |
| Template 42 | Kinetics of <gmts, gmcs=""> for <anti-rsv a="" antibody="" concentration="" igg="" neutralizing="" rsv="" titres,=""> on subjects</anti-rsv></gmts,> | |

| | with results available at all timepoints up to Day 91 <pps for="" immunogenicity="">63</pps> |
|---|---|
| Template 43 | Individual results of <anti-rsv antibody="" concentration="" igg="" neutralizing="" rsv="" titres,=""> at <day 31,61,91=""> versus prevaccination in <rsv 120="" 30,="" 60,="" mat="" rsv=""> and Placebo <pps for="" immunogenicity=""></pps></rsv></day></anti-rsv> |
| Template 44 | Geometric Mean ratios with corresponding 95% confidence interval between anti-RSV F IgG antibody concentrations and anti-RSV-A neutralising antibody titres at pre-vaccination (PPS for immunogenicity) |
| Template 45 | Geometric Mean ratios of fold increase post/pre) with corresponding 95% confidence interval between anti-RSV F IgG antibody concentrations and anti-RSV-A neutralising antibody titres at <day 31,="" 61,="" 8,="" 91="" day=""> adjusted by prevaccination ratio <pps 31,="" 61,="" 91="" <8,="" at="" day="" for="" immunogenicity="">&gt;</pps></day> |
| Template 46 | Exploratory comparisons ( <gmt, gmc=""> ratios) between RSV groups with corresponding 95% confidence interval for <anti-rsv a="" anti-rsv="" antibody="" concentration="" f="" igg="" neutralizing="" titre,=""> at Day 31 – Tukey's adjustment <pps 31="" at="" day="" for="" immunogenicity=""></pps></anti-rsv></gmt,> |
| Template 47 | Exploratory comparisons ( <gmt, gmc=""> ratios) between RSV groups with corresponding 95% confidence interval for <anti-rsv a="" anti-rsv="" antibody="" concentration="" f="" igg="" neutralizing="" titre,=""> at Day 31 <pps 31="" at="" day="" for="" immunogenicity="">66</pps></anti-rsv></gmt,> |
| Template 48 | Exploratory comparisons (Geometric mean ratios) between RSV groups with corresponding 95% confidence interval for area under curve (AUC) up to Day 91 for <anti-rsv a="" anti-rsv="" antibody="" concentration="" f="" igg="" neutralizing="" titre,=""> <pps for="" immunogenicity=""></pps></anti-rsv> |
| Template 49 | Exploratory comparisons ( <gmt, gmc=""> ratios) between RSV groups and placebo with corresponding 95% confidence interval for <rsv a="" antibody="" concentration="" f="" igg="" neutralizing="" rsv="" titre,=""> at Day 31 <pps 31="" at="" day="" for="" immunogenicity="">67</pps></rsv></gmt,> |
| Template 50 | Descriptive statistics of <anti-rsv a="" anti-rsv="" antibody="" concentration="" f="" igg="" neutralizing="" titre,="">at pre-vaccination, Day &lt;8, 31, 61, 91&gt;<pps for="" immunogenicity=""></pps></anti-rsv> |
| Template 51 | Descriptive statistics of area under the curve up to Day 91 for<br><anti-rsv a="" anti-rsv="" antibody="" antibody<br="" f="" igg="" neutralizing="" titre,="">concentration&gt; 91&gt;<pps for="" immunogenicity="">69</pps></anti-rsv> |
| Template 52 | Assessment of trend (linear or quadratic) of dose response for < <anti-rsv a="" anti-rsv="" antibody="" f="" igg<="" neutralizing="" td="" titre,=""></anti-rsv> |

| | 208068 (RSV-MAT-001)<br>Statistical Analysis Plan Final |
|---|---|
| | antibody concentration> between three RSV vaccine groups at Day 31 <pps 31="" at="" day="" for="" immunogenicity="">69</pps> |
| Template 53 | Assessment of trend (linear or quadratic) of dose response using area under curve up to Day 91 for < <anti-rsv a="" anti-rsv="" antibody="" concentration="" f="" igg="" neutralizing="" titre,=""> between three RSV vaccine groups <pps for="" immunogenicity="">70</pps></anti-rsv> |

208068 (RSV-MAT-001) Statistical Analysis Plan Final

#### **LIST OF ABBREVIATIONS**

AE Adverse event

ANCOVA Analysis of Covariance
ANOVA Analysis of Variance
CI Confidence Interval

ELISA Enzyme-linked immunosorbent assay

ES Exposed Set

GMC Geometric mean antibody concentration

GMT Geometric mean antibody titre

LL Lower Limit of the confidence interval

MedDRA Medical Dictionary for Regulatory Activities

N.A. Not Applicable

PD Protocol Deviation

PPS Per Protocol Set

SAE Serious adverse event

SAP Statistical Analysis Plan

SD Standard Deviation

SR Study Report

TFL Tables Figures and Listings

TOC Table of Content

UL Upper Limit of the confidence interval

#### 1. DOCUMENT HISTORY

| Date | Description | Protocol Version |
|-------------|---------------|------------------------------|
| 25-OCT-2018 | first version | Final Version 2- 13-AUG-2018 |

## 2. STUDY DESIGN

#### Figure 1 Study Design



- AE Adverse Events: solicited (Day 1 to Day 7); unsolicited (Day 1 to Day 30) and serious (Enrolment to Study conclusion)
- BSS Blood samples for haematology/biochemistry will be collected (~5.5 mL) from all subjects at Screening, Visit 2 (Day 8), and Visit 3 (Day 31)
- BSH Blood samples for humoral immunogenicity will be collected (~30 mL) from all subjects at Screening, Visit 2 (Day 8) Visit 3 (Day 31), Visit 4 (Day 61), and Visit 5 (Day 91)

iSRC - Internal Safety Review Committee

Contact 1- will be completed for all subjects at Day 181 (preferred contact is Phone Call)

RSV MAT 30/60/120 - RSV maternal 30/60/120µg, respectively, of the RSV maternal vaccine

Screening can occur ≤ 7 days prior to Visit 1 or on the same day, when possible

UP – Urine Pregnancy test (serum pregnancy test in country/local specific regulation) from all subjects (if Screening and Visit 1 are on the same day UP will not be repeated)

208068 (RSV-MAT-001) Statistical Analysis Plan Final

- **Experimental design**: Phase I/II, randomised, observer-blind, placebo control, multicentre study with four parallel groups
- **Duration of the study:** for each subject enrolled will be approximately 6 months from Visit 1.
  - Epoch 001: Screening Visit
  - Epoch 002: Active Vaccination phase starting at (Day 1) and concluding at, and including, Visit 3 (Day 31)
  - Epoch 003: Long Term Follow-up starting after Visit 3 (Day 31) and concluding at Contact 1 (Day181)

Any safety data collected beyond Day 31 will be collected in Epoch 003.

- **Primary Completion Date**: Visit 3 (Day 31) or last visit of Epoch 002
- Control: placebo control
- Vaccination schedule: Single intramuscular injection at Visit 1 (Day 1)
- **Treatment allocation:** Subjects will be randomised using a centralized randomisation system on internet (SBIR) at Visit 1 (Day 1). The randomisation algorithm will use a minimization procedure accounting for age (18 32 years or 33 45 years) and centre.

#### • Blinding:

Table 1 Blinding of study epochs

| Study Epochs | Blinding |
|--------------|----------------|
| 001 | N/A |
| 002 | observer-blind |
| 003 | single-blind * |

<sup>\*</sup> The study will be conducted in an observer-blind fashion through Day 91. After this day, the study will continue in a single-blind fashion.

#### • Sampling schedule

- **Blood samples for haematology/biochemistry**: will be collected (~5.5 mL) from all subjects at Screening, Visit 2 (Day 8), Visit 3 (Day 31) and any Unscheduled Visit(s).
- **Blood samples for humoral immunogenicity:** will be collected (~30 mL) from all subjects at Screening, Visit 2 (Day 8), Visit 3 (Day 31), Visit 4 (Day 61) and Visit 5 (Day 91).
- **Safety monitoring**: This study will be monitored by a blinded SRT and by an unblinded iSRC. The analyses for iSRC evaluation will be described in SAP for iSRC.

## 3. OBJECTIVES

## 3.1. Primary objective

• To evaluate the safety and reactogenicity of three dose levels (30, 60, 120 μg) of the RSV maternal investigational vaccine administered as a single intramuscular injection, as compared to placebo up to 1-month post vaccination (Day 31).

## 3.2. Secondary objective

- To evaluate the safety of three dose levels (30, 60, 120μg) of the RSV maternal investigational vaccine compared to placebo up to 6 months post vaccination (Day 181).
- To evaluate the humoral immune response to three dose levels (30, 60, 120µg) of the RSV maternal investigational vaccine compared to placebo up to 3 months post vaccination (Day 91).

## 3.3. Tertiary objective

• To further evaluate the humoral immune response to the RSV maternal vaccine.

#### 4. ENDPOINTS

## 4.1. **Primary endpoints**

- Occurrence of any adverse events (AEs) from vaccination during a 30-day follow up period, for all subjects in all groups:
  - Occurrence of each solicited local and general symptom during a 7-day follow-up period;
  - Occurrence of any unsolicited AE during a 30-day follow up period;
  - Occurrence of Serious AEs during a 30-day follow up period;
  - Occurrence of any haematological (Leukocytes, Neutrophils, Lymphocytes, Eosinophils, Haemoglobin, Platelets) and biochemical (alanine aminotransferase [ALT], aspartate aminotransferase [AST], creatinine, blood urea nitrogen [BUN]) laboratory abnormalities at Day 8 and Day 31.

# 4.2. **Secondary endpoints**

- Occurrence of SAEs from vaccination up to Day 91 and up to Day 181 for all subjects, in all groups.
- Humoral immune response to the investigational vaccine at Day 8, Day 31, Day 61 and Day 91 for all subjects in each investigational RSV vaccine groups:
  - RSV-A neutralising antibody (Nab) titres;
  - RSVPreF3 IgG antibody concentration.

## 4.3. Tertiary endpoint

Additional humoral response which may include but not limited to, RSVPreF3
specific IgG1 subclass antibody concentrations, RSV-B neutralising antibody titres,
antibody competing for binding to specific epitopes on RSVPreF3 and antibody
concentrations to residual host cell proteins in the RSVPreF3 vaccines.

## 5. ANALYSIS SETS

#### 5.1. **Definition**

Two cohorts will be defined for the purpose of the analysis: the Exposed Set (ES) and the Per-protocol set (PPS) for analysis of immunogenicity. All analyses will be performed per treatment actually administered.

## 5.1.1. Exposed Set (ES)

The ES will include all subjects with study vaccine administration documented.

- A **safety** analysis based on the ES will include all vaccinated subjects.
- An **immunogenicity** analysis based on the ES will include all vaccinated subjects for whom immunogenicity data are available.

# 5.1.2. Per-protocol set (PPS) for analysis of immunogenicity

The PPS for immunogenicity will be defined by time-point (Day 8, Day 31, Day 61 and Day 91) and will include all vaccinated subjects:

- Meeting all eligibility criteria (i.e. no protocol violation linked to the inclusion/ exclusion criteria, including age);
- Who received the study vaccine according to protocol procedures;
- Who did not receive a concomitant vaccination/medication/product leading to elimination from the PPS analysis up to the corresponding time-point as described in Section 6.6 of the protocol;
- Who did not present with an intercurrent medical condition leading to elimination from the PPS analysis up to the corresponding time-point, as described in Section 6.7 of the protocol;
- Who complied with the post-vaccination immunogenicity blood sampling schedule at the corresponding time-point, as specified in Table 2 of the SAP;
- For whom post-vaccination immunogenicity results are available for at least 1 assay at the corresponding time-point.
- The intervals allowed for the inclusion in the PPS for analysis of immunogenicity as specified in Table 2 of the SAP as bellow:

Table 2 Intervals between study visits

| | Interval | Optimal length of interval | Allowed interval for<br>PPS<br>immunogenicity |
|---|---|---|---|
| Interval to be | DOB → Visit 1 (Day 1) | 18-45 years | 18-45 years |
| considered for<br>enrollment | SCR – Visit 1 (Day 1) | 0-7 days | 0-7 days |
| Interval to be | Visit 1 (Day 1) → Visit 2 (Day 8) | 7 days | 7 - 10 days |
| considered for blood<br>sampling | Visit 1 (Day 1) $\rightarrow$ Visit 3 (Day 31) | 30 days | 30 - 45 days |
| | Visit 1 (Day 1) $\rightarrow$ Visit 4 (Day 61) | 60 days | 56 – 70 days |
| | Visit 1 (Day 1) $\rightarrow$ Visit 5 (Day 91) | 90 days | 86 - 100 days |

When presenting different time-points, the PPS for immunogenicity will be adapted for each time-point (Day 8, Day 31, Day 61 and Day 91).

# 5.2. Criteria for eliminating data from Analysis Sets

Elimination codes are used to identify subjects to be eliminated from analysis. Details are provided below for each set.

# 5.2.1. Elimination from Exposed Set (ES)

Code 1030 (Study vaccine not administered at all) and code 900 (invalid informed consent or fraud data) will be used for identifying subjects eliminated from ES.

### 5.2.2. Elimination from Per-protocol analysis Set (PPS)

## 5.2.2.1. Excluded subjects

A subject will be excluded from the PPS analysis under the following conditions:

| Code | Condition under which the code is used |
|---|---|
| 900 | Invalid informed consent or fraud data |
| 000 | (Subjects receiving a code 900 should not receive any other elimination codes) |
| 1030 | Study vaccine not administered at all |
| | (Subjects receiving a code 1030 should not receive any other elimination codes) |
| 1050 | Randomization failure (subject not randomized in the correct group) |
| | Comment: To check for manual randomisation, treatment not compatible with one assigned |
| | by SBIR |
| 1060 | Randomization code was broken |
| 1070** | Study vaccine dose not administered according to protocol |
| | Incorrect volume of the vaccine given |
| | Administration not according to protocol for reason specified by the investigator, other than |
| | side, site and route |
| | Site of the injection of vaccine is wrong or unknown |
| | Route of the study vaccine is wrong or unknown |
| | Wrong reconstitution of administered vaccine |
| 1080 | Vaccine temperature deviation |
| 1090 | Expired vaccine administered |
| 2010 | Protocol violation (inclusion/exclusion criteria including age) |
| | SCR – VIST 1 – 0-7 days# |
| | DOB – VISIT 1 – 18-45 years |

<sup>\*</sup>Attribution of these elimcodes to subject need CRDL review of individual listing

## 5.2.2.2. Right censored Data

• Data from a subject will be censored from visit x for the PPS analysis under the following conditions. The code \*\*\*\*. Vx will be used to identify subjects whose immunogenicity data should be eliminated from a specific visit onwards. For Day 8, Day 31, Day 61 and Day 91 PP, the information will be checked from vaccination up to Day 7, Day 30, Day 60 and Day 90, respectively.

<sup>\*\*</sup> Attribution of code 1070 to a subject requires CRDL confirmation

<sup>#</sup> need to be confirmed in the Pre-analysis meeting

• The code \*\*\*\*.Vx+ will also be used to identify study withdrawal.

| 1040.Vx+* | <ul> <li>Administration of concomitant vaccine(s) forbidden in the protocol</li> <li>Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine up to study completion (Contact 1 [Day 181])</li> <li>A vaccine not foreseen by the study protocol administered during 30 days following vaccination, with the exception of seasonal influenza vaccine which may be administered ≥ 15 days after the dose of study vaccine. (To note – this code will only be checked at Day 8 and Day 31 PP and will be carried forward for D61 and D91 PPS)</li> </ul> |
|---|---|
| 2040.Vx+* | <ul> <li>Administration of any medication forbidden by the protocol</li> <li>Any investigational or non-registered product (drug) other than the study vaccines used during the study period.</li> <li>Immunoglobulins and/or any blood products administered up to 90 days post study vaccination.</li> <li>Immunosuppressants or other immune-modifying drugs administered chronically (i.e. more than 14 days in total) or any long-acting immune-modifying drugs (e.g. infliximab) administered any time up to 90 days post-vaccination. For corticosteroids, this will mean ≥5mg/day prednisone or equivalent.</li> </ul> |
| 2050.Vx+* | Intercurrent medical condition Intercurrent medical condition (up to Day 91/Visit 5) that has the capability of altering immune response which may influence immune response |
| 2070.Vx+* | Concomitant infection which may influence immune response |
| 2071.Vx+ | Withdrawal from the study impacting PPS |

<sup>\*</sup>Attribution of these elimcodes to subject need CRDL review of individual listing

#### 5.2.2.3. Visit-specific censored Data

Data from visit x will be censored for the PPS analysis under the following conditions.

| Code | Condition under which the code is used |
|---|---|
| 2090.Vx | Subjects did not comply with blood sample schedule |
| | Applicable visits |
| | <ul> <li>For Day 8 PP, to check for DOSE to DAY 8 BS = 7-10 days</li> </ul> |
| | <ul> <li>For Day 31 PP, to check for DOSE to DAY 31 BS = 30-45 days</li> </ul> |
| | <ul> <li>For Day 61 PP, to check for DOSE to DAY 61 BS = 56-70 days</li> </ul> |
| | <ul> <li>For Day 91 PP, to check for DOSE to DAY 91 BS = 86-100 days</li> </ul> |
| 2100.Vx | Serological results not available post-vaccination → No immunological result at all for the specific blood sample collection timepoint Comment: - |
| | To check for availability of RSV-A neutralising antibody and/or RSVPreF3 lgG antibody result at each applicable PPS timepoint |
| 2120.Vx | Obvious incoherence or abnormality or error in immunogenicity (antibody) data*** To check on RSV-A neutralising antibody and RSVPreF3 lgG antibody result at each applicable PPS timepoint |

<sup>\*\*\*</sup> Elimination criteria for implausible RSV serum immune responses (neut and/or ELISA): More than 4-fold decrease from pre-vaccination to Day 30; After Day 30, more than 4-fold increase or more than 8 fold decrease within a 30 day period

# 5.3. Important protocol deviation not leading to elimination from per-protocol analysis set

The following important protocol deviations will be reported by groups:

- Forced randomization: In case of supplies shortage for the next assigned vaccine according to the randomization schedule at the clinical site, the randomization system will use the forced randomization procedure in order to continue to enrol and vaccinate subjects. The system moves seamlessly to the next treatment/randomization number for which vaccine supplies are available. The site will not be aware of the forced randomization event.
- Manual randomization: In case the randomization system is unavailable, the investigator has the option to request randomization to the SBIR helpdesk.
- Short follow-up: subjects who completed the last study contact before the minimum length of follow-up requirement.

#### 6. STATISTICAL ANALYSES

# 6.1. **Demography**

# 6.1.1. Analysis of demographics/baseline characteristics planned in the protocol

The analysis of demographics will be performed on the ES and on the PPS for immunogenicity.

Demographic characteristics such as age at vaccination in years, race, ethnicity, vital signs and cohort description will be summarised by group using descriptive statistics:

- Frequency tables will be generated for categorical variable such as race.
- Mean, median, standard error and range will be provided for continuous data such as age.

The distribution of subjects will be tabulated as a whole and per group and for each age category (18 - 32 years and 33 - 45 years).

Withdrawal status will be summarised by group using descriptive statistics:

- The number of subjects enrolled into the study as well as the number of subjects excluded from PPS analyses will be tabulated.
- The number of withdrawn subjects will be tabulated according to the reason for withdrawal.

#### 6.1.2. Additional considerations

- Vital signs will be presented at all time point(s) the information is collected on Exposed Set and Per Protocol Set.
- Summary of important protocol deviation leading to elimination will be presented. An individual listing will also be presented for this.
- The following table will be performed for web public disclosure
  - Percentage of Enrolled subjects by country will be tabulated by group,
  - Percentage of Enrolled subjects by age categories (18 64 years) will be tabulated by group.

# 6.2. **Exposure**

## 6.2.1. Analysis of exposure planned in the protocol

None

# 6.3. **Immunogenicity**

## 6.3.1. Analysis of immunogenicity planned in the protocol

The analysis will be performed on the applicable PPS cohort for immunogenicity and, if in any group the percentage of vaccinated subjects with serological results excluded from the PPS for analysis of immunogenicity is  $\geq 5\%$ , a second analysis will be performed on the ES.

#### 6.3.1.1. Within group assessment

Humoral Immune response to RSV vaccine

For each group, at each time point that blood samples are collected and for each assay (RSV-A NAb and RSVPreF3 IgG) (unless specified otherwise):

- GMTs/GMCs will be tabulated with 95% CI based on log-transformed values and represented graphically.
- Percentage of subjects above the sero-positivity threshold will be tabulated with exact 95% CI.
- Pre- and Post- titres/concentrations will be displayed using reverse cumulative curves.
- The distributions of RSV-A NAb titres (Percentage of subjects greater than or equal to specified thresholds (< 128, 128-256, > 256-512, > 512-1024, > 1024-2048, > 2048-4096, >4096-8192 and >8192) will be tabulated.

208068 (RSV-MAT-001) Statistical Analysis Plan Final

- Individual post-vaccination versus pre-vaccination results will be plotted using scatter plots. Results of the control group will be used as a reference.
- Geometric mean of ratios of antibody titres/concentrations post-vaccination over prevaccination will be tabulated with 95% CI.
- Distribution of the fold increase of the antibody titres (post- over pre-vaccination titers) will be tabulated.
  - Percentage of subjects with a fold increase equal to or above 2, 4, 6, 8, 10 and 12 by pre-vaccination titre category: (< 128, 128-256, > 256-512, > 512-1024, > 1024-2048, > 2048-4096, > 4096, and by cumulative category: <128, ≥128, ≥256, ≥512, ≥1024, ≥2048, ≥4096.).
- The kinetics of individual antibody titres/concentrations will be plotted as a function of time for subjects with results available at all time points.
- An analysis of variance model for repeated measures will be fitted to assess the mean profile in each group.

If deemed necessary (minimum of 10% subjects is required in both the age-category), the same analyses may be performed by age category (18 - 32 years and 33 - 45 years).

Fold increase of RSVPreF3 immunoglobulin G (IgG) antibody concentrations over fold increase of RSV-A Nab titres (Ratio of fold increase Post- over Pre-vaccination) will be tabulated using descriptive statistics. This analysis will include calculation on:

- Geometric mean ratios with corresponding 95% CIs of RSVPreF3 immunoglobulin G (IgG) antibody concentration over anti-RSV-A plaque reduction Nab titres at prevaccination for each group and
- Geometric mean ratios with corresponding 95% CIs of fold increase post/pre (Day 8, Day 31, Day 61 and Day 91/Day 1) between RSVPreF3 immunoglobulin G (IgG) antibody concentration and anti-RSV-A plaque reduction Nab titres for each group

#### 6.3.1.2. Between group assessment

Exploratory comparisons will be performed for RSV-A Nab titres and RSVPreF3 IgG antibody concentrations between the different RSV vaccine groups at Day 31. If deemed necessary, this exploratory comparison may also be done at other time-points.

- The three RSV formulations will be first compared to the Placebo in order to identify groups whose means are significantly different from the mean of the Placebo group, (alpha=2.5%, Dunnett's adjustment test for multiplicity). The model will include vaccine group as fixed effect, pre-vaccination titre/concentration. Age categories (18 - 32 years and 33 - 45 years) and/or centre will be added as the categorical covariate, if deemed necessary and is significant. For this analysis, the model will be explored and fitted via the proc mixed procedure according to the following code:

```
PROC MIXED data=sero;
CLASS subjid group age_cat center;
MODEL log_val = baseline group age_cat center
/ddfm=kenwardroger outp = pred;
Random Subjid;
lsmeans group/pdiff=control('1') adjust=dunnett cl alpha=0.05;
RUN;
```

- Estimation of GMT/GMC ratios between groups with corresponding 95% CI using an ANCOVA model on the logarithm10 transformation of the titres/concentrations. This model includes:
  - The vaccine group as the fixed effect
  - The pre-vaccination titre/concentration as the covariate
  - Age groups (18 32 years and 33 45 years) and/or centre as the categorical covariate if deemed necessary
- Linear and quadratic trend of dose response will be tested using appropriate contrasts.

For the between group analysis among groups and trend tests, the model will be explored and fitted via the proc mixed procedure according to the following code:

```
PROC MIXED data=sero;
CLASS subjid group age_cat center;
MODEL log_val = baseline group age_cat center
/ddfm=kenwardroger outp = pred;
Random Subjid;
lsmeans group/pdiff, cl alpha=0.05;
ods output diffs = diff lsmeans = lsm covparms=cov;
Contrast 'Linear' group 0 -4 -1 5;
Contrast 'Quadratic' group 0 -3 1 2;
RUN:
```

## 6.3.2. Additional considerations

Few points have been added as additional consideration: -

- The immune analysis at Day 31 for Step 1 subject will only be performed on Exposed Set.
- Summary statistics of RSV-A Nab titres and RSVPreF3 IgG concentration (Minimum, Mean, median, SD, 1<sup>st</sup> quartile, 3<sup>rd</sup> quartile, Maximum) will be presented.
- The thresholds for presentation of titres in distribution table and for fold increase will be further adjusted at Day 91 analysis as needed.
- Area under curve (AUC) for each individual will be calculated using linear trapezoid method on titres/concentrations up to 91 days as data permit and summary statistics will be presented. Following loge-transformation, AUC will be analyzed by analysis of covariance (ANCOVA) fitting baseline as covariate and vaccine group as a fixed effect. Point estimates and associated 95% confidence intervals for the group difference will be constructed using the residual error term. These point estimates and associated 95% confidence intervals will then be exponentially back-transformed to provide point estimates and 95% confidence intervals for ratio on fold change. Trend of dose response will also be explored using AUC. The program for the analysis will be similar to between group analysis among vaccine groups and trend tests at day 31. The AUC will be calculated as

$$AUC = \sum_{i=2}^{n} \frac{1}{2} (m_{i-1} - m_i) * (t_{i-1} - t_i)$$

where  $m_i$  corresponds to the  $i^{th}$  measurement and  $t_i$  corresponds to the  $i^{th}$  time point. Each subject's rectangular areas must be added together to estimate the AUC.

- Only subjects having at least 3 post vaccination immune results will be considered for AUC calculation.
- An analysis of variance model for repeated measures will be fitted to assess the mean profile in each group over time.

```
PROC MIXED data=sero;
CLASS subjid group visit age_cat center;
   MODEL log_val = baseline group | visit age_cat
center/ddfm=kenwardroger outp = pred;
   Random Subjid;
lsmeans group*visit/pdiff, cl alpha=0.05;
ods output diffs = diff lsmeans = lsm covparms=cov;
RUN;
```

## 6.4. **Analysis of safety**

## 6.4.1. Analysis of safety planned in the protocol

The analysis of safety will be performed on the ES.

### 6.4.1.1. Within group analysis

The percentage of subjects with at least one **local AE** (solicited and unsolicited), with at least one **general AE** (solicited and unsolicited) and with any AE during the 7-day or 30-day follow-up period after vaccination will be tabulated with exact 95% CI. The same computations will be done for any ≥ Grade 2 AEs, for any AEs considered related to vaccination, for any Grade 3 AEs considered related to vaccination and for AEs resulting in medically attended visit.

The percentage of subjects reporting each individual **solicited local AE** (any, each grade, resulting in medically attended visit) during the 7-day follow-up period after vaccination will also be tabulated based on maximum intensity per subject for each study vaccine group. The percentage of subjects reporting each individual **solicited general AE** (any, each grade, any related, any Grade 2 related, any Grade 3 related, resulting in medically attended visit) during the 7-day follow-up period after vaccination will also be based on maximum intensity per subject for each study vaccine group.

For fever during the 7-day follow-up period after vaccination, the number and percentage of subjects reporting any fever and fever by half degree (°C) cumulative increments will be reported. Similar tabulations will be performed for causally related fever, Grade 3 causally related fever and fever resulting in a medically attended visit. In addition, the prevalence of any and Grade 3 fever will be presented graphically over time after vaccination.

The percentage of subjects with any **unsolicited** symptoms within 30 days after vaccination with its exact 95% CI will be tabulated by group and by MedDRA System Organ Class and preferred term. Similar tabulation will be done for Grade 3 unsolicited symptoms, for any causally related unsolicited symptoms, for Grade 3 causally related unsolicited symptoms and for unsolicited symptoms resulting in a medically attended visit (the verbatim reports of unsolicited symptoms will be reviewed by a physician and the signs and symptoms will be coded according to the MedDRA Dictionary for Adverse Reaction Terminology. Every verbatim term will be matched with the appropriate Preferred Term).

**SAEs** reported throughout the study will be described in detail.

**Pregnancy** exposures throughout the study and pregnancy outcomes will be described in detail (if applicable).

208068 (RSV-MAT-001) Statistical Analysis Plan Final

The percentage of subjects using **concomitant medication** (any medication, any antipyretic and any antipyretic taken prophylactically, respectively) during the 7-day follow-up period (Day 1 - 7), 30 days follow-up (Day 1 - 30), between Day 1 - Day 91 and between Day 1- Day 181 after vaccination, will be summarized by group.

For all subjects in each group and each **haematology and biochemistry** parameter:

- The percentage of subjects having haematology and biochemistry results below or above the local laboratory normal ranges will be tabulated for each time point.
- The maximum grading post-vaccination (up to Day 8 and up to Day 31) versus baseline (Screening) and the percentage of subjects with laboratory parameters above or equal to Grade 1, Grade 2, Grade 3 and Grade 4 will be tabulated (Grades will be based on the FDA Guidance for Industry "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials", see Table 4 and Table 5: FDA toxicity grading scale. Those laboratory parameters not included on FDA Toxicity Grading Scale will not be graded).

#### 6.4.2. Additional considerations

The percentage of subjects with at least one grade 3 **local AE** (solicited and unsolicited), with at least one grade 3 **general AE** (solicited and unsolicited) and with any grade 3 AE during the 7-day or 30-day follow-up period after vaccination will be tabulated with exact 95% CI.

Descriptive summary of the number of days with solicited local/general adverse event during the 7 day (Days 1-7) post-vaccination period will be presented.

The percentage of subjects with SAE within 30 days (Day 1-30) after vaccination with its exact 95% CI will be tabulated by group and by MedDRA preferred term. Similar table will be generated for SAE from study start up to Day 90 and from study start up to study end.

SAEs, death, and withdrawal due to AE(s) reported during the entire study will be tabulated.

#### 6.4.2.1. Exclusion of implausible solicited Adverse Event

Some local and systemic adverse events will be directly measured by the subject and will be subject to a reconciliation process, even if they are biologically implausible. Therefore, these implausible measurements will be removed from the analysis but included in listings. Implausible measurements are summarized in the table below:

Table 3 Implausible Solicited Adverse Events

| Parameter | Implausible measurements |
|------------------|----------------------------------|
| Body temperature | ≤ 33°C or ≥ 42°C |
| Erythema | Measurements < 0 mm |
| | For subjects ≥ 6 years: ≥ 900 mm |
| Swelling | Measurements < 0 mm |
| | For subjects ≥ 6 years: ≥ 500 mm |

#### 6.4.2.2. Combined Solicited and Unsolicited Adverse Events

A summary of subjects with all combined solicited (regardless of their duration) and unsolicited adverse events will be provided. Solicited adverse events will be coded by MedDRA as per the following codes

| Solicited symptom | Lower level term code | Corresponding Lower level term decode |
|---|---|---|
| Pain | Injection site pain | 10022086 |
| Redness | Redness at injection site | 10022098 |
| Swelling | Swelling at injection site | 10053425 |
| Fatigue | Fatigue | 10016256 |
| Fever | Fever | 10016558 |
| Headache | Headache | 10019211 |
| Gastrointestinal symptoms | Gastrointestinal disorder | 10017944 |

Please note - to check for AE term in cDISC during dry run

For clintrial.gov and EudraCT posting purposes, a summary of combined solicited and unsolicited non-serious adverse events will be produced by System Organ Class and preferred terms and according to occurrence of each event.

#### 7. ANALYSIS INTERPRETATION

All comparative analyses will be descriptive with the aim to characterise the difference in immunogenicity between groups. These descriptive analyses should be interpreted with caution considering that there is no adjustment for multiplicity for most of these comparisons.

## 8. CONDUCT OF ANALYSES

## 8.1. Sequence of analyses

In order to obtain early immunogenicity data of the different formulations of the investigational RSV Maternal vaccine, an interim analysis will be performed on Exposed Set when immunogenicity data up to Day 31 for the Step 1 subjects becomes available. This analysis will be performed on Exposed Set on data as available (i.e partially clean or non-clean data). The templates and listings to be reported for this analysis will be detailed in TFL TOC of this SAP.

To ensure the study team remains blinded, the analysis will be performed by an unblinded statistician outside GSK and the iSRC will act as a firewall team, to review the aggregated summaries for risk of unblinding of individual subjects, before these are released to the team. For this analysis only a statistical report will be prepared

The final statistical analyses will be performed in 2 steps:

- A first analysis will be performed when all safety and immunogenicity data up to at least Day 91 is available in all subjects. At this point, the study statistician will be unblinded (i.e. will have access to the individual subject treatment assignments), but no individual listings will be provided to investigators until the final study report. However, summary results may lead to the unblinding of some specific subjects in case an event occurred only in one group; steps will be taken to minimize this risk.
- The final analysis covering all primary and secondary endpoints as well as any evaluated tertiary endpoint(s) will be performed when all data up to study conclusion are available. A clinical study report will only be written at this stage and individual listings will be provided as part of it.

If the data for tertiary endpoints becomes available at a later stage, (an) additional analysis/analyses will be performed. These data will be documented in annex(es) to the study report and will be made available to the investigators at that time

208068 (RSV-MAT-001) Statistical Analysis Plan Final

| Description | Analysis<br>ID | Disclosure Purpose (CTRS=public posting, SR=study report, internal) | Dry run<br>review<br>needed (Y/N) | Study Headline Summary (SHS)requiring expedited communication to upper management (Yes/No) | Reference for TFL |
|---|---|---|---|---|---|
| Final - Up to Day<br>181 | E1_01 | CTRS, Study report | Y | Y | See sheet<br>TOC-DAY181<br>in TFL TOC |
| D31-Step 1 | E1_02 | Internal | Y | Y | See sheet<br>TOC-S1-D31 in<br>TFL TOC |
| Up to Day 91 | E1_03 | CTRS | Y | Y | See sheet<br>TOC-DAY91 in<br>TFL TOC |

# 8.2. Statistical considerations for interim analyses

All analyses are descriptive. Therefore, the conduct of interim analyses has no impact on interpretation of study results.

### 9. CHANGES FROM PLANNED ANALYSES

None

# 10. LIST OF FINAL REPORT TABLES, LISTINGS AND FIGURES

The TFL TOC provides the list of tables/listings and figures needed for the study report. It also identifies the tables eligible for each analyses and their role (synopsis, in-text, post-text, SHS, CTRS,...). Note that all TFL aimed to be included as post-text are noted as post-text even if these are tabulation of individual data such as listing of SAE. The post-text material contains all source material for the study report and accordingly a post-text table may be redundant with an in-text table.

The following group names will be used in the TFLs, to be in line with the T-domains:

| Group order in tables | Group label in tables | Group definition for footnote |
|---|---|---|
| 1 | RSV MAT 30 | Subject receiving RSVPreF3 low dose |
| 2 | RSV MAT 60 | Subject receiving RSVPreF3 mid dose |
| 3 | RSV MAT 120 | Subject receiving RSVPreF3 high dose |
| 4 | Placebo | Subject receiving placebo |

The following sub-group names will be used in the TFLs

| Sub-group order in tables | Sub-group label in tables | Sub-group definition for footnote |
|---|---|---|
| 1 | 18-32Y | Subjects 18-32 years of age |
| 2 | 33-45Y | Subjects 33-45 years of age |

# 11. ANNEX 1 STANDARD DATA DERIVATION RULE AND STATISTICAL METHODS

#### 11.1. Statistical Method References

The exact two-sided 95% CIs for a proportion within a group will be the Clopper-Pearson exact CI [Clopper CJ, Pearson ES. The use of confidence or fiducial limits illustrated in the case of binomial. *Biometrika*. 1934;26:404-413].

#### 11.2. Standard data derivation

#### 11.2.1. Date derivation

- SAS date derived from a character date: In case day is missing, 15 is used. In case day & month are missing, 30June of the year will be used.
- Onset day for an event (AE, medication, etc.): The onset day is the number of days between the study vaccination and the onset/start date of the event. This is 1 for an event starting on the same day as a vaccination. See SAS date derived in case the start date of the event is incomplete.
- Duration: Duration of an event is expressed in days. It is the number of days between the start & the stop dates + 1. Therefore, duration is 1 day for an event starting & ending on the same day.

# 11.2.2. Demography

- For computation of age, following rules need to be considered:
  - Age will be calculated as the number of years between the date of birth and the date of first vaccination.
  - To ensure that the collection of date of birth will not jeopardise the privacy of Personally Identifiable Information (PII), only a partial date of birth (MMYYYY or YYYY as per local regulation) will be collected.
  - Note that due to incomplete date, the derived age may be incorrect by 1 year when month is missing from the birthdate. This may lead to apparent inconsistency between the derived age and the eligibility criteria/the age category used for randomization.

208068 (RSV-MAT-001) Statistical Analysis Plan Final

- For the summary of vital sign, the descriptive statistics will be presented in:
  - Height in cm
  - Weight in kg
  - BMI in kg/m2
  - Temperature in celsius
  - Heart rate in beats per minute
  - Respiratory rate in breaths per minute
  - Systolic and Diastolic Blood pressure in mmHg
- Conversion of weight to kg The following conversion rule is used:
  - Weight in Kilogram= weight in Pounds / 2.2

The result is rounded to 2 decimals.

- Conversion of height to cm The following conversion rule is used:
  - Height in Centimetres = Height in Inch \* 2.54

The result is rounded to the unit (ie no decimal).

- Conversion of temperature to °C The following conversion rule is used:
  - Temperature in °Celsius = ((Temperature in °Fahrenheit -32) \*5)/9

The result is rounded to 1 decimal.

# 11.2.3. Immunogenicity

- For a given subject and given immunogenicity measurement, missing or nonevaluable measurements will not be replaced. Therefore, an analysis will exclude subjects with missing or non-evaluable measurements.
  - For the within-group assessment, the descriptive analysis performed for each assay at each timepoint will exclude subjects with a missing or non-evaluable measurement.
  - For the between group assessments, the Analysis of covariance (ANCOVA) model will be fitted at each timepoint based on the subjects having a result at both the baseline and the considered timepoint.
- The Geometric Mean Concentrations/Titres (GMC/Ts) calculations are performed by taking the anti-log of the mean of the log titre transformations. Antibody titres below the cut-off of the assay will be given an arbitrary value of half the cut-off of the assay for the purpose of GMC/T calculation. The cut-off value will be defined by the laboratory before the analysis.

208068 (RSV-MAT-001) Statistical Analysis Plan Final

- The 95% CI for GMT will be obtained within each group separately. The 95% CI for the mean of log-transformed titre will be first obtained assuming that log-transformed titres were normally distributed with unknown variance. The 95% CI for the GMT will then be obtained by exponential transformation of the 95% CI for the mean of the log-transformed titres.
- A seronegative subject is a subject whose antibody titre is below the cut-off value of the assay. A seropositive subject is a subject whose antibody titre is greater than or equal to the cut-off value of the assay.
- GMT/GMC ratios will be obtained using an ANCOVA model on the logarithm-transformed titres. The ANCOVA model will include the vaccine group as fixed effect, pre-vaccination titre as covariate and age groups (18 32 years and 33 45 years) and/or centre as the categorical covariate if deemed necessary. GMT/GMC ratios and their CI (based on Tukey multiple adjustment) will be derived as exponential-transformation of the corresponding group contrast in the model.
- The CI for GMT ratio will be obtained by exponential-transformation of the CI for the group least square mean of the log-transformed titres/concentration of the above ANCOVA model. Confidence intervals adjusted for multiple testing or other kind of significance adjustment will be produced.
- All CI computed will be two-sided 95% CI.

### 11.2.4. Safety

- For a given subject and the analysis of solicited symptoms within 7 days post-vaccination, missing or non-evaluable measurements will not be replaced. Therefore, the analysis of the solicited symptoms based on the Exposed Set will include only vaccinated subjects with documented safety data (i.e., symptom screen completed). More specifically the following rules will be used:
  - Subjects who documented the absence of a solicited symptom after vaccination will be considered not having that symptom after vaccination.
  - When a specific symptom is marked as having occurred following a specific vaccination (i.e. SDTM CE.CEOCCUR=Y for the specified post-vaccination period for the symptom in question), any missing daily recordings will be given imputed values to allow them to contribute to the 'Any' rows but not to specific grade rows of the symptom summary tables.
  - Dose without symptom sheets documented will be excluded.
- For analysis of unsolicited adverse events, such as serious adverse events or adverse
  events by primary MedDRA term, and for the analysis of concomitant medications,
  all vaccinated subjects will be considered. Subjects who did not report the event or
  the concomitant medication will be considered as subjects without the event or the
  concomitant medication respectively.

Note that for all tables described in this section, the way the percentage of subjects will be derived will depend on the event analysed (see table below for details). As a result, the N value will differ from one table to another.

| Event | N used for deriving % per subject for Vaccination phase |
|---|---|
| Concomitant vaccination | All subjects with study vaccine administered |
| Solicited general symptom | All subjects with at least one solicited general symptom documented as either present or absent (i.e., symptom screen completed) |
| Solicited local symptom Unsolicited symptom | All subjects with at least one solicited local symptom documented as either present or absent (i.e., symptom screen completed) All subjects with study vaccine administered |
| Concomitant medication | All subjects with study vaccine administered |

# 11.2.5. Number of decimals displayed:

The following decimal description from the decision rules will be used for the demography, immunogenicity and safety/reactogenicity.

| Display Table | Parameters | Number of decimal digits |
|---|---|---|
| Demographic characteristics | Mean, median age | 1 |
| Demographic characteristics | SD (age) | 1 |
| Immunogenicity | Ratio of GMT/C | 2 |
| All summaries | % of difference, including LL & UL of CI | 2 |
| All summaries | p-value | 3 |

# 12. ANNEX 2: TOXICITYGRADING SCALE FOR LABORATORY ASSESSMENTS

Table 4 FDA toxicity grading scales for biochemistry parameters

| Serum* | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially Life<br>Threatening<br>(Grade 4)** |
|---|---|---|---|---|
| Creatinine – mg/dL | 1.5 – 1.7 | 1.8 – 2.0 | 2.1 – 2.5 | > 2.5 or requires dialysis |
| Blood Urea Nitrogen BUN mg/dL | 23 – 26 | 27 – 31 | > 31 | Requires<br>dialysis |
| Liver Function Tests -ALT, AST increase by factor | 1.1 – 2.5 x ULN | 2.6 – 5.0 x ULN | 5.1 – 10 x ULN | > 10 x ULN |

ULN = upper limit of the normal range.

<sup>\*</sup> The laboratory values provided in the tables serve as guidelines and are dependent upon institutional normal parameters. Institutional normal reference ranges should be provided to demonstrate that they are appropriate.

<sup>\*\*</sup> The clinical signs or symptoms associated with laboratory abnormalities might result in characterization of the laboratory abnormalities as Potentially Life Threatening (Grade 4). For example, a low sodium value that falls within a Grade 3 parameter (125-129 mE/L) should be recorded as a Grade 4 hyponatremia event if the subject had a new seizure associated with the low sodium value.

Table 5 FDA toxicity grading scales for hematology parameters

| Hematology* | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially<br>Life<br>Threatening<br>(Grade 4) |
|---|---|---|---|---|
| Hemoglobin (Female) - gm/dL | 11.0 – 12.0 | 9.5 – 10.9 | 8.0 – 9.4 | < 8.0 |
| Hemoglobin (Female)<br>change from baseline value -<br>gm/dL | Any decrease -<br>1.5 | 1.6 – 2.0 | 2.1 – 5.0 | > 5.0 |
| WBC Increase - cell/mm3 | 10 800 – 15 000 | 15 001 – 20 000 | 20 001 – 25 000 | > 25 000 |
| WBC Decrease - cell/mm3 | 2 500 – 3 500 | 1 500 – 2 499 | 1 000 – 1 499 | < 1 000 |
| Lymphocytes Decrease - cell/mm3 | 750 – 1 000 | 500 – 749 | 250 – 499 | < 250 |
| Neutrophils Decrease - cell/mm3 | 1 500 – 2 000 | 1 000 – 1 499 | 500 – 999 | < 500 |
| Eosinophils - cell/mm3 | 650 – 1 500 | 1 501 - 5 000 | > 5 000 | Hypereosino philic |
| Platelets Decreased - cell/mm3 | 125 000 –<br>140 000 | 100 000 –<br>124 000 | 25 000 – 99 000 | < 25 000 |

<sup>\*</sup> The laboratory values provided in the tables serve as guidelines and are dependent upon institutional normal parameters. Institutional normal reference ranges should be provided to demonstrate that they are appropriate.

## 13. ANNEX 3: STUDY SPECIFIC MOCK TFL

The data display, title and footnote are for illustration purpose and will be adapted to the study specificity as indicated in the TFL TOC. Note that there may be few changes between the study specific SAP mock TFL and the final TFLs as editorial/minor changes do not require a SAP amendment.

## 13.1. List of individual data listing

Appendix Table I.A - Elimination codes

Appendix Table I.Ai – Important Protocol deviations

Appendix Table I.B – Demography

Appendix Table IBii - Physical examination/vital signs

Appendix Table I.Ci - Dates of birth, Informed consent, Vaccination and blood sampling, Contact

Appendix Table I.Cii - Reason for visit not done

Appendix Table I.D - General medical history - Physical examination

Appendix Table I.Ei – Study Conclusion

Appendix Table I.Eii – Screening conclusion

Appendix Table I.G / I.H - Vaccination procedure

208068 (RSV-MAT-001) Statistical Analysis Plan Final

Appendix Table I.I - Reason for not administration of vaccine

Appendix Table I.J - Reason for non-eligibility

Appendix Table II.Ai - Solicited local adverse events

Appendix Table II.B - Solicited general adverse events

Appendix Table II.Ci - Unsolicited adverse events within (30) days post-vaccination

Appendix Table II.Cii - Unsolicited adverse events after (30) days post-vaccination

Appendix Table II.Di - Concomitant medications

Appendix Table II.Dii - Concomitant vaccinations

Appendix Table III.A – Immunogenicity

Appendix Table IV.A – Haematology and Biochemistry

Appendix Table V.A – Pregnancy report

## 13.2. Template of Tables and Figures

#### Template 1 Number of subjects by country and center <Exposed Set>

| | | | <each group=""> <eac<br>N=XXXX N=XX</eac<br></each> | | h group><br>(XX | Total<br>N=XXXX | |
|---|---|---|---|---|---|---|---|
| Country | Center | n | % | n | % | n | % |
| <each country=""></each> | <each center=""></each> | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| | All | XXX | XX.X | XXX | XX.X | XXX | XX.X |

#### <each group>:

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

n = number of subjects in a given center or country

N = total number of subjects

 $% = n/N \times 100$ 

Center = GSK Biologicals assigned center number

# Template 2 Number of subjects vaccinated, completed and withdrawn with reason for withdrawal – up to <Day 31, Day 91, study end> <Exposed set>

| | <each group=""><br/>N=XXXX</each> | | Total<br>N=XXXX | |
|---|---|---|---|---|
| | n | % | n | % |
| Number of subjects vaccinated | XXX | | XXX | XXX |
| End of study status | | | | |
| [EACH CATEGORY] | XXX | | XXX | xxx |
| Reasons for withdrawal: | | | | |
| [REASONS] | XXX | | XXX | XXX |

#### <each group>:

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

Vaccinated = number/percentage of subjects who were vaccinated in the study

Completed = number/percentage of subjects who completed last study visit

Withdrawn = number/percentage of subjects who did not perform the last study visit

Unknown = number/percentage of subjects who have not come for the last visit yet

Template 3 Visit attendance – up to <Day 31, Day 91, study end> <Exposed set>

| | | <each group=""> N=XXX</each> | |
|---|---|---|---|
| Visit | Status | n | % |
| <each visit=""></each> | Attended | | |
| | Not attended yet | | |
| | Permanent discontinuation prior to or at this visit | | |
| | Not attended | | |
| CONCLUSION | Completed | | |

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

N = Number of subjects in each group or in total

n/% = number / percentage of subjects in a given category

Conclusion = date of last study visit or withdrawal

208068 (RSV-MAT-001) Statistical Analysis Plan Final

Template 4 Summary of important protocol deviation leading to elimination from Per protocol set <Enrolled Set>

| | Ea | Each group<br>N= | | Total<br>N= |
|---|---|---|---|---|
| Title | n | % | n | % |
| At least one Important Protocol Deviation | | | | |
| Assessment or time point completion | | | | |
| Missed assessment | | | | |
| Out of window assessment for | | | | |
| immunogenicity | | | | |
| Eligibility Criteria Not Met | | | | |
| Inclusion Exclusion Criteria Not Met | | | | |
| Excluded medication, vaccine or device | | | | |
| Medication, excluded by the protocol, was administered | | | | |
| Vaccine, excluded by the protocol, was administered | | | | |
| Intercurrent medical conditions | | | | |
| Developed intercurrent medical condition leading to PPS | | | | |
| exclusion | | | | |
| Fraudulent Data | | | | |
| Fraudulent Data | | | | |
| Informed Consent | | | | |
| Informed consent not signed and/or dated by subject | | | | |
| Study procedures | | | | |
| Randomization procedures | | | | |
| Wrong study treatment/administration/dose | | | | |
| Not administering any study treatment | | | | |
| Study treatment not administered per | | | | |
| protocol | | | | |
| Essential serological data missing | | | | |
| Obvious incoherence or abnormality or error in data | | | | |

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

N = Number of subjects in each group or in total

Occ = number of occurrences = number of important protocol deviations

n/% = number / percentage of subjects with important protocol deviations

Template 5 Consort flow - Part 1 from enrolment to randomization <All Enrolled Set>

| | Total<br>N= | |
|--------------------------------------------------------|-------------|-----|
| | n | % |
| NUMBER OF SUBJECTS ELIMINATED PRIOR TO RANDOMIZATION | | |
| Consent Withdrawal, Not Due To A Serious Adverse Event | | |
| Consent Withdrawal, Not Due To An Adverse Event | 2 | 0.3 |
| Eligibility Criteria Not Fulfilled | | |
| Lost To Follow-Up | | |
| Migrated / Moved From The Study Area | | |
| Missing | | |
| Other | | |
| NUMBER OF SUBJECTS INCLUDED IN RANDOMIZED SET | | |

N = Number of subjects

n = Number of subjects enrolled by site

% = n / Number of subjects with available results x100

All Enrolled Set includes Screen Failures and non-Randomized subjects

Withdrawal reason "Other" corresponds to Subject Enrollment target reached before Randomization
208068 (RSV-MAT-001) Statistical Analysis Plan Final

Template 6 Consort – Part II from randomization to exposure for each study group <AII Randomised Set>

| group van Kandonnood oor | | | |
|---|---|---|---|
| | Each group<br>N= | Total<br>N= | |
| | | n | % |
| NUMBER OF SUBJECTS ELIMINATED PRIOR TO EXPOSURE | | | |
| Consent Withdrawal, Not Due To A Serious Adverse Event | | | |
| Consent Withdrawal, Not Due To An Adverse Event | | 2 | 0.3 |
| Eligibility Criteria Not Fulfilled | | | |
| Lost To Follow-Up | | | |
| Migrated / Moved From The Study Area | | | |
| NUMBER OF SUBJECTS INCLUDED IN EXPOSED SET | | | |

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

N = Number of subjects

n = Number of subjects randomised by site

% = n / Number of subjects with available results x 100

Template 7 Consort flow - Part 3 from exposure to per protocol set, per study group <Exposed Set>

| | Each group<br>N= | | | otal<br>I= |
|---|---|---|---|---|
| | n | % | n | % |
| NUMBER OF SUBJECTS ELIMINATED FROM PER PROTOCOL SET AT | | | | |
| DAY <8, 31, 61, 91> | | | | |
| ELIMINATIONS | | | | |
| Eligibility Criteria Not Met (2010) | | | | |
| Missed Assessment (2100) | | | | |
| Out Of Window Treatment Administration (2080) | | | | |
| Study Treatment Not Administered Per Protocol (1070) | | | | |
| WITHDRAWALS | | | | |
| Consent Withdrawal, Not Due To An Adverse Event | | | | |
| Lost To Follow-Up | | | | |
| Serious Adverse Event | | | | |
| NUMBER OF SUBJECTS INCLUDED IN PER PROTOCOL SET AT DAY | | | | |
| <8, 31, 61, 91> | | | | |

N = Number of subjects

n = Number of subjects enrolled by site

<sup>% =</sup> n / Number of subjects with available results x 100

208068 (RSV-MAT-001) Statistical Analysis Plan Final

### Template 8 Summary of demographic characteristics <Exposed set, PPS for immunogenicity at Day <8, 31, 61, 91>>

| | <each group=""> N=XXXX</each> | | <each group=""> N=XXXX</each> | | | otal<br>XXXX |
|---|---|---|---|---|---|---|
| | Value or n | % | Value or n | % | Value or n | % |
| Age in years at <timepoint></timepoint> | | | | | | |
| N with data | XXX | | xxx | | xxx | |
| Mean | XXX.X | | xxx.x | | XXX.X | |
| SD | XXX.X | | xxx.x | | xxx.x | |
| Median | XXX.X | | xxx.x | | xxx.x | |
| Minimum | XXX | | xxx | | XXX | |
| Maximum | XXX | | xxx | | XXX | |
| Age category at (vaccination) | | | | | | |
| 18-32 years | xxx | XX.X | xxx | XX.X | XXX | XX.X |
| 33-64 years | xxx | XX.X | xxx | XX.X | XXX | XX.X |
| Ethnicity | | | | | | |
| <each ethnicity=""></each> | xxx | XX.X | xxx | XX.X | XXX | XX.X |
| | XXX | XX.X | xxx | XX.X | xxx | XX.X |
| Geographic Ancestry | | | | | | |
| <each ancestry="" geographic=""></each> | XXX | XX.X | xxx | XX.X | xxx | XX.X |
| | XXX | XX.X | xxx | XX.X | XXX | XX.X |

#### <each group>:

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

N = total number of subjects

n/% = number / percentage of subjects in a given category

Value = value of the considered parameter

N with data = number of subjects with documentation of the corresponding data

SD = standard deviation

208068 (RSV-MAT-001) Statistical Analysis Plan Final

## Template 9 Summary of vital signs characteristics <Exposed set, PPS for immunogenicity at Day <8, 31, 61, 91>>

| | | | <each group=""> N =</each> | Total<br>N = |
|---|---|---|---|---|
| Visit | Characteristics | Parameters | Value | Value |
| Each visit> | Height (Cm) | N with data | | |
| | 9(**) | Mean | | |
| | | SD | | |
| | | Median | | |
| | | Minimum | | |
| | | Maximum | | |
| | Weight (Kg) | N with data | | |
| | Weight (Ng) | Mean | | |
| | | SD | | |
| | | Median | | |
| | | Minimum | | |
| | | Maximum | | |
| | BMI | N with data | | |
| | DIVII | | | |
| | | Mean | | |
| | | SD | | |
| | | Median | | |
| | | Minimum | | |
| | | Maximum | | |
| | Heart rate (Beats per minute) | N with data | | |
| | | Mean | | |
| | | SD | | |
| | | Median | | |
| | | Minimum | | |
| | | Maximum | | |
| | Respiratory rate (Breaths per minute) | N with data | | |
| | | Mean | | |
| | | SD | | |
| | | Median | | |
| | | Minimum | | |
| | | Maximum | | |
| | Temperature/(Oral) (°C) | N with data | | |
| | , | Mean | | |
| | | SD | | |
| | | Median | | |
| | | Minimum | | |
| | | Maximum | | |
| | Systolic Blood pressure (mmHg) | N with data | | |
| | Cystolic Blood pressure (Illilling) | Mean | | |
| | | SD | | |
| | | Median | | |
| | | Minimum | | |
| | Diagtalia Diagdanas / | Maximum | | |
| | Diastolic Blood pressure (mmHg) | N with data | | |
| | | Mean | | |
| | | SD | | |
| | | Median | | |
| | | Minimum | | $\perp$ |
| | | Maximum | | |

<each group>:

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose
RSV MAT 120 = Subject receiving RSVPreF3 high dose
Placebo = Subject receiving placebo
N = total number of subjects
N with data = number of subjects with documentation of the corresponding data
Value = value of the considered parameter
SD = standard deviation

Template 10 Deviations from specifications for age and intervals between study visits <Exposed Set>

| | | | <each group=""></each> | | <each group<="" th=""><th>&gt;</th></each> | > |
|---|---|---|---|---|---|---|
| | Interval | | | | | |
| Type of interval | range | | Value or n | % | Value or n | % |
| Age | 18 - 45 years | N | xxx | | XXX | |
| | | n | xxx | xx.x | xxx | xx.x |
| | | Minimum | xxx | | XXX | |
| | | Maximum | xxx | | XXX | |
| SCR – VISIT 1 | 0 – 7 Days | N | xxx | | XXX | |
| | | n | xxx | XX.X | xxx | XX.X |
| | | Minimum | xxx | | XXX | |
| | | Maximum | xxx | | XXX | |
| /ISIT 1 – VISIT 2 | 7 – 10 Days | N | xxx | | xxx | |
| | | n | xxx | XX.X | XXX | XX.X |
| | | Minimum | xxx | | XXX | |
| | | Maximum | xxx | | XXX | |
| /ISIT 1 – VISIT 3 | 30 – 45 Days | N | xxx | | XXX | |
| | | n | xxx | XX.X | XXX | XX.X |
| | | Minimum | xxx | | XXX | |
| | | Maximum | xxx | | XXX | |
| /ISIT 1 – VISIT 4 | 56 – 70 Days | N | xxx | | XXX | |
| | | n | xxx | XX.X | XXX | XX.X |
| | | Minimum | xxx | | XXX | |
| | | Maximum | xxx | | XXX | |
| /ISIT 1 – VISIT 5 | 86 – 100<br>Days | N | xxx | | xxx | |
| | | n | xxx | xx.x | XXX | xx.x |
| | | Minimum | xxx | | XXX | |
| | | Maximum | xxx | | XXX | |
| /ISIT 1 – PHC 1 | 165 – 195<br>Days | N | xxx | | xxx | |
| | , | n | XXX | XX.X | xxx | xx.x |
| | | Minimum | XXX | | xxx | |
| | | Maximum | xxx | | xxx | |

#### <each group (pooled groups)>:

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

N = total number of subjects with available results

n/% = number / percentage of subjects with results outside of the interval

range = minimum-maximum for age and intervals

#### Template 11 Study Population – Up to <Day 91, study end> <Exposed Set>

| | <each group=""> N=XXXX</each> | <each group=""> N=XXXX</each> | Total<br>N=XXXX |
|---|---|---|---|
| Number of subjects | | | |
| Planned, N | XXX | XXX | XXX |
| Randomised, N <cohort name=""></cohort> | XXX | XXX | XXX |
| Completed, n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| <unknown></unknown> | XXX | XXX | XXX |
| Demographics | | | |
| N <cohort name=""></cohort> | XXX | XXX | XXX |
| Females:Males | XXX:XXX | XXX:XXX | XXX:XXX |
| Mean Age, <unit> (SD)</unit> | xxx.x (xxx.x) | xxx.x (xxx.x) | xxx.x (xxx.x) |
| Median Age, <unit> (minimum, maximum)</unit> | xxx (xxx,xxx) | xxx (xxx,xxx) | xxx (xxx,xxx) |
| <most category="" frequent="" of="" race=""></most> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| <second category="" frequent="" most="" of="" race=""></second> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| <third category="" frequent="" most="" of="" race=""></third> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

#### <each group>:

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

N = Total number of subjects

SD = Standard deviation

#### Template 12 Number of enrolled subjects by country

| | <each group=""><br/>N =</each> | Total<br>N = |
|-----------------|--------------------------------|--------------|
| Characteristics | n | n |
| Country | | |

#### <each group>:

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

N = Number of enrolled subjects

n= number of enrolled subjects included in each group or in total for a given country or for all countries

#### Template 13 Number of enrolled subjects by age category

| | | <each group=""><br/>N =</each> | Total<br>N = |
|---|---|---|---|
| Characteristics | Categories | n | n |
| Age category | Adults [18-45 years] | | |
| | Missing | | |

#### <each group>:

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

N = Number of enrolled subjects

n= number of enrolled subjects included in each group or in total for a given age category or for all age categories Missing = age at study vaccination unknown

#### Template 14 Minimum and maximum activity dates <Exposed set>

| | | <each group=""></each> | <each group=""></each> | Overall |
|---|---|---|---|---|
| Visit | Parameter | Date | Date | Date |
| Description | | | | |
| <inform consent=""></inform> | Minimum | | | |
| | Maximum | | | |
| [Randomisatio n] | Minimum | | | |
| | Maximum | | | |
| <each visit=""></each> | Minimum | | | |
| | Maximum | | | |

#### <each group>:

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

Template 15 Compliance in completing solicited symptoms information <Exposed Set>

| | <each group=""></each> | | | | <each group=""></each> | |
|---|---|---|---|---|---|---|
| Symptom information | N | n | Compliance (%) | N | n | Compliance (%) |
| General SS | | | | | | |
| Local SS | | | | | | |

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

N=Number of administered doses

n = number of doses with SS returned

General SS = Symptom screens used for the collection of general solicited AEs

Local SS = Symptom screens used for the collection of local solicited AEs

Compliance (%) =  $(n / N) \times 100$ 

Template 16 Incidence and nature of <any, grade 2 and 3, grade 3, related, grade 3 related, > adverse events (unsolicited and solicited) <requiring medical attention> reported during the <7,30>-days (Day 1-<7,30>) post-vaccination period <Exposed Set>

| | <each group=""></each> | | | | <each group=""></each> | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | _ | | 95% CI | | | 95% CI | | | | |
| Symptoms | N | n | % | LL | UL | N | n | % | LL | UL |
| Any symptom | | | | | | | | | | |
| General symptoms | | | | | | | | | | |
| Local symptoms | | | | | | | | | | |

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

N = number of subjects with the administered dose

n/% = number/percentage of subjects presenting at least one type of symptom

95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

208068 (RSV-MAT-001) Statistical Analysis Plan Final

## Template 17 Incidence of solicited local adverse events reported during the 7-day (Days 1-7) post-vaccination period by maximum grading <Exposed Set>

| | | <each group=""></each> | | | | |
|---|---|---|---|---|---|---|
| | | | | | | 95 % CI |
| Symptom | Туре | N | n | % | LL | UL |
| Pain | All | | | | | |
| | Grade 1 | | | | | |
| | Grade 2 | | | | | |
| | Grade 3 | | | | | |
| | Medical advice | | | | | |
| | Onset ≤48h | | | | | |
| Redness (mm) | All | | | | | |
| , , | >20 - ≤50 | | | | | |
| | >50 - ≤100 | | | | | |
| | >100 | | | | | |
| | Medical advice | | | | | |
| | Onset ≤48h | | | | | |
| Swelling (mm) | All | | | | | |
| | >20 - ≤50 | | | | | |
| | >50 - ≤100 | | | | | |
| | >100 | | | | | |
| | Medical advice | | | | | |
| | Onset ≤48h | | | | | |

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

N = number of subjects with the documented dose

n/% = number/percentage of subjects reporting the type of symptoms as maximum intensity during the follow-up

CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

The maximum intensity of local injection site redness/swelling was coded as follows:

- 1: >20 mm to  $\leq$  50 mm
- $2: > 50 \text{ mm to} \le 100 \text{ mm}$
- 3: > 100 mm

Please note - to check for AE term in cDISC during dry run

208068 (RSV-MAT-001) Statistical Analysis Plan Final

### Template 18 Number of days with solicited local adverse event during the 7-day (Days 1-7) post-vaccination period <Exposed Set>

| | | <each group=""></each> | <each group=""></each> |
|---|---|---|---|
| Symptom | Statistic | value | value |
| Pain | n | XXXX | XXXX |
| | Mean | XX.X | XX.X |
| | Minimum | XX.X | XX.X |
| | Q1 | XX.X | XX.X |
| | Median | XX.X | XX.X |
| | Q3 | XX.X | XX.X |
| | Maximum | XX.X | XX.X |
| Redness (mm) | n | XXXX | XXXX |
| | Mean | XX.X | XX.X |
| | Minimum | XX.X | XX.X |
| | Q1 | XX.X | XX.X |
| | Median | XX.X | XX.X |
| | Q3 | XX.X | XX.X |
| | Maximum | XX.X | XX.X |
| Swelling (mm) | n | XXXX | XXXX |
| | Mean | XX.X | XX.X |
| | Minimum | XX.X | XX.X |
| | Q1 | XX.X | XX.X |
| | Median | XX.X | XX.X |
| | Q3 | XX.X | XX.X |
| | Maximum | XX.X | XX.X |

#### <each group>:

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

n = number of doses with the symptom

Q1 = 25th percentile

Q3 = 75th percentile

Please note – to check for AE term in cDISC during dry run

Template 19 Percentage of subjects reporting solicited local adverse events (any grade /grade 2,3/ grade 3) during the 7-day (Days 1-7) post-vaccination period by maximum intensity <Exposed set>



RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

Please note – to check for AE term in cDISC during dry run

#### Template 20 Incidence of solicited general adverse event reported during the 7day (Days 1-7) post-vaccination period by maximum grading <Exposed Set>

| | | Each | | gro | oup |
|----------------------------|-----------------|------|-----|-----|------|
| | | | | 95 | % CI |
| Symptom | Туре | ı | 1 % | LL | UL |
| Fatigue | All | | | | |
| · · | Grade 1 | | | | |
| | Grade 2 | | | | |
| | Grade 3 | | | | |
| | Related | | | | |
| | Grade 2 Related | | | | |
| | Grade 3 Related | | | | |
| | Medical advice | | | | |
| | Onset ≤48h | | | | |
| Gastrointestinal | All | | | | |
| symptoms | | | | | |
| , . | Grade 1 | | | | |
| | Grade 2 | | | | |
| | Grade 3 | | | | |
| | Related | | | | |
| | Grade 2 Related | | | | |
| | Grade 3 Related | | | | |
| | Medical advice | | | | |
| | Onset ≤48h | | | | |
| Headache | All | | | | |
| | Grade 1 | | | | |
| | Grade 2 | | | | |
| | Grade 3 | | | | |
| | Related | | | | |
| | Grade 2 Related | | | | 1 |
| | Grade 3 Related | | | | |
| | Medical advice | | | | - |
| | Onset ≤48h | | | | |
| Temperature/(Oral)<br>(°C) | All | | | | |
| ( - / | ≥38.0 | | | | |
| | >38.5 | | | | |
| | >39.0 | | | | 1 |
| | >39.5 | | | | |
| | >40.0 | | | | 1 |
| | Related | | | | 1 |
| | >38.5 Related | t | 1 | | + |
| | >39.0 Related | | | | + |
| | >39.5 Related | 1 | 1 | | + |
| | >40.0 Related | 1 | | | 1 |
| | Medical advice | + | + | | + |
| | Onset ≤48h | 1 | | | 1 |

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

N = number of subjects with the documented dose

n/% = number/percentage of subjects reporting the type of symptom as maximum intensity during the follow-up period 95%CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

All=any grade>0 for Fatigue, Gastrointestinal symptoms, Headache and any ≥38.0°C for Temperature

208068 (RSV-MAT-001) Statistical Analysis Plan Final

Related\*= any grade>0 for Fatigue, Gastrointestinal symptoms, Headache and any  $\geq$ 38.0°C for Temperature considered related to vaccination by the investigator

Please note – to check for AE term in cDISC during dry run

Template 21 Number of days with solicited general adverse event during the 7-day (Days 1-7) post-vaccination period <Exposed Set>

| | | <each group=""></each> | <each group=""></each> |
|---|---|---|---|
| Symptom | Statistic | value | value |
| atigue | n | xxxx | XXXX |
| | Mean | XX.X | XX.X |
| | Minimum | XX.X | XX.X |
| | Q1 | XX.X | XX.X |
| | Median | XX.X | XX.X |
| | Q3 | XX.X | XX.X |
| | Maximum | XX.X | XX.X |
| Sastrointestinal | n | XXXX | XXXX |
| ymptoms | Mean | XX.X | XX.X |
| | Minimum | XX.X | XX.X |
| | Q1 | XX.X | XX.X |
| | Median | XX.X | XX.X |
| | Q3 | XX.X | XX.X |
| | Maximum | XX.X | XX.X |
| leadache | n | XXXX | XXXX |
| | Mean | XX.X | XX.X |
| | Minimum | XX.X | XX.X |
| | Q1 | XX.X | XX.X |
| | Median | XX.X | XX.X |
| | Q3 | XX.X | XX.X |
| | Maximum | XX.X | XX.X |
| emperature (Oral) (°C) | n | XXXX | XXXX |
| | Mean | XX.X | XX.X |
| | Minimum | XX.X | XX.X |
| | Q1 | XX.X | XX.X |
| | Median | XX.X | XX.X |
| | Q3 | XX.X | XX.X |
| | Maximum | XX.X | XX.X |

#### <each group>:

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

n = number of doses with the symptom

Q1 = 25th percentile

Q3 = 75th percentile

Please note – to check for AE term in cDISC during dry run

Template 22 Percentage of subjects reporting fever (any and grade 3) and other solicited general adverse events (any grade /grade 2,3/ grade 3) during the 7-day (Days 1-7) post-vaccination period by maximum intensity <Exposed set>



RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

Grade 3 fever = Temperature >39.0 °C

Please note – to check for AE term in cDISC during dry run

208068 (RSV-MAT-001) Statistical Analysis Plan Final

Template 23 Percentage of subjects reporting the occurrence of <any, grade 3> <unsolicited symptoms, serious adverse events> classified by MedDRA Primary System Organ Class and Preferred Term <with causal relationship to vaccination, with medically attended visit>, within the 30-day (Days 1-30) post-vaccination period <Exposed Set>

| | | Eac<br>N = | h gı | rou | ) | |
|---|---|---|---|---|---|---|
| | | | | | | 5%<br>CI |
| Primary System Organ Class (CODE) | Preferred Term (CODE) | n* | n | % | LL | UL |
| At least one symptom | | | | | | |
| Gastrointestinal disorders (10017947) | Diarrhoea (10012735) | | | | | |
| · | Teething (10043183) | | | | | |
| | Vomiting (10047700) | | | | | |
| General disorders and administration site conditions (10018065) | Pyrexia (10037660) | | | | | |
| Immune system disorders (10021428) | Seasonal allergy (10048908) | | | | | |
| Infections and infestations (10021881) | Conjunctivitis (10010741) | | | | | |
| , , | Otitis media (10033078) | | | | | |
| | Paronychia (10034016) | | | | | |
| | Tonsillitis (10044008) | | | | | |
| | Tonsillitis streptococcal (10044013) | | | | | |
| | Viral upper respiratory tract infection | | | | | |
| | (10047482) | | | | | |
| Injury, poisoning and procedural complications (10022117) | Arthropod bite (10003399) | | | | | |
| | Face injury (10050392) | | | | | |
| | Head injury (10019196) | | | | | |
| Skin and subcutaneous tissue disorders (10040785) | Miliaria (10027627) | | | | | |

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = = number of subjects included in the considered analysis set in each group

n\* = number of events reported

n/% = number/percentage of subjects reporting the symptom at least once

95% CI = exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

n\* will only be generated for the CTRS posting

# Template 24 Percentage of subjects reporting the occurrence of <serious adverse events> classified by MedDRA Primary System Organ Class and Preferred Term from <vaccination up to Day 91 visit, from vaccination up to study end> <Exposed Set>

| • | · | | acł<br>I = | n gr | oup |
|---|---|---|---|---|---|
| | | | | | 5%<br>CI |
| Primary System Organ Class (CODE) | Preferred Term (CODE) | n | % | LL | UL |
| At least one symptom | | | | | |
| Gastrointestinal disorders (10017947) | Diarrhoea (10012735) | | | | |
| | Teething (10043183) | | | | |
| | Vomiting (10047700) | | | | |
| General disorders and administration site conditions (10018065) | Pyrexia (10037660) | | | | |
| Immune system disorders (10021428) | Seasonal allergy (10048908) | | | | |
| Infections and infestations (10021881) | Conjunctivitis (10010741) | | | | |
| | Otitis media (10033078) | | | | |
| | Paronychia (10034016) | | | | |
| | Tonsillitis (10044008) | | | | |
| | Tonsillitis streptococcal (10044013) | | | | |
| | Viral upper respiratory tract infection (10047482) | | | | |
| Injury, poisoning and procedural complications (10022117) | Arthropod bite (10003399) | | | | |
| , | Face injury (10050392) | | | | |
| | Head injury (10019196) | | | | |
| Skin and subcutaneous tissue disorders (10040785) | Miliaria (10027627) | | | | |

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects included in the considered cohort in each group

n/% = number/percentage of subjects reporting the symptom at least once

95% CI = exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

Template 25 Number and percentage of subjects taking a concomitant medication <during the <7,30>- day (Days 1-<7,30>) post-vaccination period, from vaccination to Day 91 visit/study end> <Exposed Set>

| • | | <each group=""></each> | | | |
|---|---|---|---|---|---|
| | | | | 9 | 95% CI |
| Туре | N | n | % | LL | UL |
| Any | | | | | |
| Any antipyretics | | | | | |
| Prophylactic antipyretics | | | | | |

#### <each group>:

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

N = total number of subjects with the administered dose

n/% = number/percentage of subjects took the specified type of concomitant medication at least once during the considered period

95%CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

208068 (RSV-MAT-001) Statistical Analysis Plan Final

## Template 26 Distribution of change from baseline in hematology and biochemistry with respect to normal laboratory ranges <Exposed Set>

| | | | | | | group |
|---|---|---|---|---|---|---|
| Laboratory parameter | Timing | Range<br>indicator at<br>Baseline<br>(SCR) | Range indicator at timing | N | n | % |
| Alanine<br>Aminotransferase | PI(D8) | Unknown | Unknown | | | |
| | | | Below | | | |
| | | | Within | | | |
| | | | Above | | | |
| | | Below | Unknown | | | |
| | | | Below | | | |
| | | | Within | | | |
| | | | Above | | | |
| | | Within | Unknown | | | |
| | | | Below | | | |
| | | | Within | | | |
| | | | Above | | | |
| | | Above | Unknown | | | |
| | | | Below | | | |
| | | | Within | | | |
| | | | Above | | | |
| | PI (D31) | | | | | |
| Aspartate<br>Aminotransferase | | | | | | |
| Creatinine | | | | | | |
| Blood Urea Nitrogen | | | | | | |
| Hemoglobin | | | | | | |
| Leukocytes (White<br>Blood Cells) | | | | | | |
| Neutrophil | | 1 | | | | |
| Eosinophil | | | | | | |
| Platelets | | | | | | |
| . 10.0.00 | | | 1 | <u> </u> | | 1 |

#### <each group>:

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

N = number of subjects with available results for the specified laboratory parameter and timing in a given baseline category

n/% = number/percentage of subjects in the specified category

Below = below the normal laboratory range defined for the specified laboratory parameter

Within = within the normal laboratory range defined for the specified laboratory parameter

Above = above the normal laboratory range defined for the specified laboratory parameter

SCR= Screening

PI (D8): Post-vaccination at Day 8

PI (D31): Post-vaccination at Day 31

Template 27 Summary of hematology and biochemistry results by maximum grade up to <VISIT 2 (D8), VISIT 3 (D31)> post vaccination versus baseline <Exposed Set>

| | | | <eac< th=""><th>ch gro</th><th>oup &gt;</th></eac<> | ch gro | oup > |
|---|---|---|---|---|---|
| Laboratory parameter | Baseline<br>(SCR) | Visit 2 to<br>Visit X | N | n | % |
| Alanine Aminotransferase(ALT) | Unknown | Unknown | | | |
| | | Grade 0 | | | |
| | | Grade 1 | | | |
| | | Grade 2 | | | |
| | | Grade 3 | | | |
| | | Grade 4 | | | |
| | Grade 0 | | | | |
| | Grade 1 | | | | |
| | Grade 2 | | | | |
| | Total | | | | |
| Aspartate | | | | | |
| Aminotransferase(AST) | | | | | |
| Creatinine | | | | | |
| Eosinophils increase | | | | | |
| Hemoglobin decrease | | | | | |
| Lymphocytes decrease | | | | | |
| Neutrophil (decrease) | | | | | |
| Platelet count decrease | | | | | |
| White Blood Cells (WBC) | | | | | |
| decrease | | | | | |
| White Blood Cells (WBC) | | | | | |
| increase | | | | | |

#### <each group>:

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

N = number of subjects with at least one available result for the specified laboratory parameter and follow-up period n/% = number/percentage of subjects reporting at least once the laboratory event when the maximum grading over the follow-up period is considered

SCR=Screening

Template 28 Summary of haematology change from baseline by maximum grade in the specified category <up to VISIT2 (D8), up to VISIT 3 (D31) ><Exposed set>

| | | | | | | | MAT 120 | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | I | | N = | | N = | | N = | N = | | | 1 = |
| Laboratory parameter | Maximum grade | n | % | n | % | n | % | n | % | n | % |
| Hemoglobin (Change from baseline) | Other | | | | | | | | | | |
| | Grade 2 | | | | | | | | | | |
| | Grade 3 | | | | | | | | | | |
| | Grade 4 | | | | | | | | | | |

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

N = number of subjects with at least one available result for the specified laboratory parameter and follow-up period % = percentage of subjects reporting at least once the laboratory event when the maximum grading over the follow-up period is considered

% = n / Number of subjects with available results x 100

Other=all Unknown, Grade 0 and Grade 1

208068 (RSV-MAT-001) Statistical Analysis Plan Final



Note: This figure is just a template.

Template 30 Solicited and unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 1-30) post-vaccination period including number of events - SAE excluded <Exposed Set>

| | | <eac< th=""><th>up&gt;</th></eac<> | up> | |
|---|---|---|---|---|
| Primary System Organ Class (CODE) | Preferred Term (CODE) | n* | n | % |
| At least one symptom | | | | |
| <each soc=""></each> | <each pt="" term=""></each> | | | |

#### <each group>:

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with the administered dose

n\* = number of events reported

n/% = number/percentage of subjects reporting the symptom at least once

208068 (RSV-MAT-001) Statistical Analysis Plan Final

Template 31 Number (%) of subjects with serious adverse events including number of events reported <within 30 days (Days 1-30) post vaccination period><from vaccination up to Day 91 visit, Study end> <Exposed Set>

| | | | <each group=""> N =</each> | | |
|---|---|---|---|---|---|
| Type of Event | Primary System Organ Class | Preferred Term (CODE) | n* | n | % |
| SAE | At least one symptom | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | |
| Related SAE | At least one symptom | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | |
| Fatal SAE | At least one symptom | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | |
| Related fatal SAE | At least one symptom | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | |

#### <each group>:

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

N = number of subjects with the administered dose

n\* = number of events reported

n/% = number/percentage of subjects reporting the symptom at least once

208068 (RSV-MAT-001) Statistical Analysis Plan Final

### Template 32 Listing of all SAEs <within 30 day (Days 1-30) post-vaccination period, from vaccination up to <Day 91, study end> ><Exposed Set>

| Gr | oup | Sub.<br>No. | Sex | Country | Race | Age at<br>onset<br>(Year) | Preferred<br>term | Primary<br>System<br>Organ<br>Class | MED<br>type | Dose | Day of onset | Duration | Intensity | Causality | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

Please note that this table will be presented on group blinded during Day 91 analysis.

### Template 33 Listing of adverse events, SAEs and solicited symptoms leading to withdrawal from the study <within 30 days (Days 1-30) post-vaccination period><during vaccination up to <Day 91, study end> <Exposed Set>

| Group | Subject No. | Country | Race | AE D | escrip) | tion | SAE | Causality | Outcome | Type of discontinuation |
|---|---|---|---|---|---|---|---|---|---|---|

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

Please note that this table will be presented on group blinded during Day 91 analysis.

25-OCT-2018 Page 55 of 70

208068 (RSV-MAT-001) Statistical Analysis Plan Final

Template 34 Listing of all pregnancies from vaccination up to study end <Exposed Set>

| Gro | IP Sub.<br>No. | Country | • | <br> | _ , | outcome | Gestational weeks at birth/miscarriage /termination |
|---|---|---|---|---|---|---|---|

RSV MAT 30 = Subject receiving RSV PreF3 low dose RSV MAT 60 = Subject receiving RSV PreF3 mid dose RSV MAT 120 = Subject receiving RSV PreF3 high dose

Placebo = Subject receiving placebo

25-OCT-2018 Page 56 of 70

208068 (RSV-MAT-001) Statistical Analysis Plan Final

# Template 35 Number and percentage of subjects with <RSV-A neutralising antibody titre, RSV IgG antibody concentration> equal to or above <cut-off> and <GMTs/GMCs> <PPS for immunogenicity, Exposed Set>

| | | | | | ≥cut- | off ur | nit | ( | GMT/GMC | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | 95 | % CI | | 95 | % CI | | |
| Antibody | Group | Timing | N | n | % | LL | UL | value | LL | UL | Min | Max |
| <rsv-a<br>NAb, RSV<br/>IgG<br/>antibody&gt;</rsv-a<br> | <each<br>group&gt;</each<br> | PRE | | | | | | | | | | |
| • | | PI(D8) | | | | | | | | | | |
| | | PI(D31) | | | | | | | | | | |
| | | PI(D61) | | | | | | | | | | |
| | | PI(D91) | | | | | | | | | | |

#### <each group>:

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

GMT/GMC = geometric mean antibody titre/concentration calculated on all subjects

N = Number of subjects with available results

n/% = number/percentage of subjects with titre equal to or above specified value

95% CI = 95% confidence interval; LL = lower limit, UL = upper limit

MIN/MAX = Minimum/Maximum

PRE= Pre-vaccination at screening

PI(D8) = Post-vaccination at Day 8

PI(D31) = Post-vaccination at Day 31

PI(D61) = Post-vaccination at Day 61

PI(D91) = Post-vaccination at Day 91

To check for the disclosure name for the antibody for 1st column of the table

### Template 36 Distribution of RSV-A neutralising antibody titre <PPS for immunogenicity <at Day X>>

| | | | Each group | | |
|---|---|---|---|---|---|
| Antibody | Timing | Titre | N | n | % |
| RSV-A NAb | <pre><pre, pi(d31),="" pi(d61),="" pi(d8),="" pi(d91)=""></pre,></pre> | <128 | | | |
| | , , | ≥128 | | | |
| | | ≥256 | | | |
| | | ≥512 | | | |
| | | ≥1024 | | | |
| | | ≥2048 | | | |
| | | ≥4098 | | | |

#### <each group>:

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

N = number of subjects with available results

n/% = number/percentage of subjects with titre within the specified criterion

PRE= Pre-vaccination at screening

PI(D8) = Post-vaccination at Day 8

PI(D31) = Post-vaccination at Day 31

PI(D61) = Post-vaccination at Day 61

PI(D91) = Post-vaccination at Day 91

Please note that the categories of the titre presentation are not fixed and will be adjusted at time of D91 analysis

Template 37 Distribution of fold of anti-RSV-A neutralising antibody titre by prevaccination titre category <PPS for immunogenicity>

| | | | | | Eac<br>rou |
|---|---|---|---|---|---|
| change RSV-A NAb <1 <128 P ≥128-≤256 >256-≤512 >1024-≤2048 >2048-≤4096 >4096 Total ≥1 - <2 ≥2 ≥4 ≥6 ≥8 ≥8 | Timing | N | n | % | |
| RSV-A NAb | | <128 | PI(D8)<br>PI(D31) | | |
| | PI(D3'<br>PI(D6'<br>≥128-≤256 | r I(D01) | | | |
| | | >256-≤512 | | | |
| | | >1024-≤2048 | | | |
| | | >2048-≤4096 | | | |
| | | >4096 | | | |
| | | Total | | | |
| | dy change Fold change Pre-vaccination status Timing N n N n % NAb <1 | | | | |
| | ≥2 | | | | |
| | change /-A NAb <1 | | | | |
| | ≥6 | | | | |
| | ≥8 | Sold Pre-vaccination status Timing N n % | | | |
| | ≥10 | Fold change | | | |
| | ≥12 | | | | |

<each group>:

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

208068 (RSV-MAT-001) Statistical Analysis Plan Final

N = number of subjects with pre- and corresponding post-vaccination results available n/% = number/percentage of subjects with titre fold change meeting the specified criterion

PI(D8) = Post-vaccination at Day 8

PI(D31) = Post-vaccination at Day 31

PI(D61) = Post-vaccination at Day 61

PI(D91) = Post-vaccination at Day 91

Please note that the categories of the titre presentation are not fixed and will be adjusted at time of D91 analysis

Template 38 Geometric mean of the individual ratio of <RSV-A neutralizing antibody titres, RSV IgG antibody concentrations> at <Day 8, Day 31, Day 61, Day 91> compared to pre-vaccination with 95% CI <PPS for immunogenicity<at Day 31>>

| | | | <gmt,< th=""><th>C&gt; rati</th><th>0</th><th></th></gmt,<> | C> rati | 0 | |
|---|---|---|---|---|---|---|
| | | | | | 95% | <b>6 CI</b> |
| Group | Time point description | Time point description | Ratio order | Value | LL | UL |
| RSV MAT 30 | PI(D31) | PRE | PI(D31) / PRE | | | |
| RSV MAT 60 | PI(D31) | PRE | PI(D31) / PRE | | | |
| RSV MAT<br>120 | PI(D31) | PRE | PI(D31) / PRE | | | |
| Placebo | PI(D31) | PRE | PI(D31) / PRE | | | |

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

<GMT,C> = geometric mean antibody <titres, concentration> calculated on all subjects

N = Number of subjects with available results at the two considered time points

95% CI = 95% confidence interval; LL = lower limit, UL = upper limit

PRE= Pre-vaccination at screening

PI(D8) = Post-vaccination at Day 8

PI(D31) = Post-vaccination at Day 31

PI(D61) = Post-vaccination at Day 61

PI(D91) = Post-vaccination at Day 91

## Template 39 Estimated <GMTs,GMCs> and 95% CIs for <RSV-A neutralising antibody titre, RSV IgG antibody concentration> (PPS for immunogenicity)

| | | | | Estima | ted | GMT |
|---|---|---|---|---|---|---|
| | | | | | 959 | % CI |
| Antibody | Group | Timing | Ν | Value | LL | UL |
| <rsv-a antibody="" concentration="" igg="" nab,="" rsv=""></rsv-a> | RSV MAT 30 | PRE | | | | |
| | | PI(D8) | | | | |
| | | PI(D31) | | | | |
| | | PI(D61) | | | | |
| | | PI(D91) | | | | |
| | RSV MAT 60 | PRE | | | | |
| | | PI(D8) | | | | |
| | | PI(D31) | | | | |
| | | PI(D61) | | | | |
| | | PI(D91) | | | | |
| | RSV MAT 120 | PRE | | | | |
| | | PI(D8) | | | | |
| | Placebo PRE | | | | | |
| | | PI(D8) | | | | |

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

GMT/C = geometric mean for <anti-RSV A Neutralizing antibody titre, RSV IgG antibody concentration> estimated by the ANOVA model for repeated measures

N = Number of subjects with available results

95% CI = 95% confidence interval (ANOVA model); LL = lower limit, UL = upper limit

PRE= Pre-vaccination at screening

PI(D8) = Post-vaccination at Day 8

PI(D31) = Post-vaccination at Day 31

PI(D61) = Post-vaccination at Day 61

PI(D91) = Post-vaccination at Day 91

Template 40 <GMTs, GMCs> and their 95% CIs for <RSV-A neutralising antibody titres, RSV IgG antibody concentration> at each timepoint up to Day <31,91> <PPS for immunogenicity>



RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

<GMT,C> = geometric mean antibody <titre, concentration> calculated on all subjects

95% CI = 95% confidence interval

PRE = Pre-vaccination at screening

PI(D8) = Post-vaccination at Day 8

PI(D31) = Post-vaccination at Day 31

PI(D61) = Post-vaccination at Day 61

PI(D91) = Post-vaccination at Day 91

Note: This graph is provided as an example. For each assay separately, this graph will display the 4 groups and the 5 immuno timepoints: PRE, PI(D8), PI(D31), PI(D61) and PI(D91)

Template 41 Reverse cumulative distribution curves for <anti-RSV-A neutralising antibody titres, RSV IgG antibody concentrations> in each group at pre-vaccination and <Day 8, Day 31, Day 61, Day 91> <PPS for immunogenicity>



cut-off = 8.00 Anti-RSV A Neutralizing Antibody

antibody fiter titres (EL.U/ml)

RSV MAT 30 = Subject receiving RSVPreF3 low dose RSV MAT 60 = Subject receiving RSVPreF3 mid dose RSV MAT 120 = Subject receiving RSVPreF3 high dose Placebo = Subject receiving placebo

Template 42 Kinetics of <GMTs, GMCs> for <anti-RSV A neutralizing antibody titres, RSV IgG antibody concentration> on subjects with results available at all timepoints up to Day 91 <PPS for immunogenicity>



RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

Please note that graph is provided as example (our groups and timepoints are different)

Template 43 Individual results of <anti-RSV neutralizing antibody titres, RSV IgG antibody concentration> at <Day 31,61,91> versus pre-vaccination in <RSV MAT 30, RSV MAT 60, RSV MAT 120> and Placebo <PPS for immunogenicity>



RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

Figure is only a template. Actual will be done for the assays mentioned in the titles and for each group.

Template 44 Geometric Mean ratios with corresponding 95% confidence interval between anti-RSV F IgG antibody concentrations and anti-RSV-A neutralising antibody titres at pre-vaccination (PPS for immunogenicity)

| | | | | | | | | | GM ratio | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | % CI | | 95% CI | | | 95% | 6 CI |
| Timing | Group description | N | IgG Total<br>GMC | LL | UL | RSV-A neut<br>GMT | LL | UL | Value | LL | UL |
| PRE | <each group=""></each> | | | | | | | | | | |
| PRE | | | | | | | | | | | |
| PRE | | | | | | | | | | | |
| PRE | | | | | | | | | | | |

#### <each group>:

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

N = Number of subjects with available results at pre-vaccination for IgG antibody concentration and RSV-A neutralizing antibody

GMC = Geometric mean antibody concentration calculated on all subjects for anti-RSV F IgG antibody concentration

GMT = Geometric mean antibody titre calculated on all subjects for RSV-A neutralizing antibody titres

GM Ratio=Geometric mean of individual ratio of IgG antibody concentration to RSV-A neutralizing antibody titre for each group

95% CI = 95% confidence interval; LL = lower limit, UL = upper limit

PRE = Pre-vaccination at screening

Template 45 Geometric Mean ratios of fold increase post/pre) with corresponding 95% confidence interval between anti-RSV F IgG antibody concentrations and anti-RSV-A neutralising antibody titres at <Day 8, Day 31, Day 61, Day 91> adjusted by pre-vaccination ratio <PPS for immunogenicity at Day <8, 31, 61, 91>>

| | | | | | | | | | GN | IF Rat | tio |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | 95 | % CI |
| Timepoint | Group | N | IgG Total | 95% ( | Cl | RSV-A neut | 95% | | Value | LL | UL |
| - | _ | | GMF | LL | UL | GMF | LL | UL | | | |
| PI(D31) | <each group=""></each> | | | | | | | | | | |
| PI(D61 | | | | | | | | | | | |
| PI(D91) | | | | | | | | | | | |

#### <each group>:

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

N = Number of subjects with available results at the two considered time points for IgG antibody concentration and anti-RSV-A neutralizing antibody titres

GMF = Geometric mean of fold increase post over pre-vaccination

GMF Ratio= Geometric mean of individual ratio of fold increase for each group

95% CI = 95% confidence interval; LL = lower limit, UL = upper limit

PRE = Pre-vaccination at screening

PI(D8) = Post-vaccination at Day 8

PI(D31) = Post-vaccination at Day 31

PI(D61) = Post-vaccination at Day 61

PI(D91) = Post-vaccination at Day 91

Template 46 Exploratory comparisons (<GMT, GMC> ratios) between RSV groups with corresponding 95% confidence interval for <anti-RSV A neutralizing antibody titre, anti-RSV F IgG antibody concentration> at Day 31 – Tukey's adjustment <PPS for immunogenicity at Day 31>

| | | | | | GN | IT ratio | | |
|---|---|---|---|---|---|---|---|---|
| | | | | | | | | key's<br>% Cl |
| Antibody | Group<br>description | N Adjusted<br><gmt,<br>GMC&gt;</gmt,<br> | Group<br>description | N Adjusted<br><gmt,<br>GMC&gt;</gmt,<br> | Ratio order | Value | LL | UL |
| <anti-rsv a="" antibody="" antibody,="" igg="" neutralizing="" rsv=""> PI(D8)</anti-rsv> | RSV MAT<br>120 | | RSV MAT 30 | | RSV MAT<br>120/RSV<br>MAT 30 | | | |
| ` ' | RSV MAT<br>120 | | RSV MAT 60 | | RSV MAT<br>120/ RSV<br>MAT 60 | | | |
| | RSV MAT 60 | | RSV MAT 30 | | RSV MAT<br>60/RSV MAT<br>30 | | | |

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Adjusted GMT = geometric mean antibody titre adjusted for age cat, center and baseline titre

N = Number of subjects with both pre- and post-vaccination results available

Tukey's 95% CI = 95% confidence interval for the GMT/GMC ratio (ANCOVA model: adjustment for age\_cat, center and baseline titre - pooled variance; Tukey's adjustment), LL = lower limit, UL = upper limit

Age\_cat is 1 for subject within age interval of 18-32 years and 2 for 33-45 years

PI(D31) = Post-vaccination at Day 31

Template 47 Exploratory comparisons (<GMT, GMC> ratios) between RSV groups with corresponding 95% confidence interval for <anti-RSV A neutralizing antibody titre, anti-RSV F IgG antibody concentration> at Day 31 <PPS for immunogenicity at Day 31>

| | | | | | | | GMT | ratio | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | 95<br>CI | % |
| Antibody | Group<br>description | N | Adjusted<br><gmt,<br>GMC&gt;</gmt,<br> | Group<br>description | N | Adjusted<br><gmt,<br>GMC&gt;</gmt,<br> | Ratio order | Value | LL | . UL |
| <anti-rsv a<br="">Neutralizing Antibody,<br/>RSV IgG antibody&gt;<br/>PI(D8)</anti-rsv> | RSV MAT<br>120 | | | RSV MAT 30 | | | RSV MAT<br>120/RSV MAT<br>30 | | | |
| , | RSV MAT<br>120 | | | RSV MAT 60 | | | RSV MAT<br>120/ RSV<br>MAT 60 | | | |
| | RSV MAT 60 | | | RSV MAT 30 | | | RSV MAT<br>60/RSV MAT<br>30 | | | |

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Adjusted GMT = geometric mean antibody titre adjusted for age cat, center and baseline titre

N = Number of subjects with both pre- and post-vaccination results available

95% CI = 95% confidence interval for the GMT/GMC ratio (ANCOVA model: adjustment for age\_cat, center and baseline titre - pooled variance), LL = lower limit, UL = upper limit

Age\_cat is 1 for subject within age interval of 18-32 years and 2 for 33-45 years

PI(D31) = Post-vaccination at Day 31

Template 48 Exploratory comparisons (Geometric mean ratios) between RSV groups with corresponding 95% confidence interval for area under curve (AUC) up to Day 91 for <anti-RSV A neutralizing antibody titre, anti-RSV F IgG antibody concentration> <PPS for immunogenicity>

| | | | | | | | GM r | atio | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | 95°<br>CI | % |
| Antibody | Group description | N | Adjusted<br><gm></gm> | Group description | N | Adjusted<br><gm></gm> | Ratio order | Value | LL | UL |
| <anti-rsv a="" neutralizing<br="">Antibody, RSV IgG<br/>antibody&gt;<br/>PI(D8)</anti-rsv> | RSV MAT 120 | | | RSV MAT 30 | | | RSV MAT<br>120/RSV MAT<br>30 | | | |
| | RSV MAT 120 | | | RSV MAT 60 | | | RSV MAT 120/<br>RSV MAT 60 | | | |
| | RSV MAT 60 | | | RSV MAT 30 | | | RSV MAT<br>60/RSV MAT<br>30 | | | |

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Adjusted GM = geometric mean of area under curve (AUC) adjusted for age\_cat, center and baseline titre N = Number of subjects with both pre- and post-vaccination results available

95% CI = 95% confidence interval for the GMT/GMC ratio (ANCOVA model: adjustment for age\_cat, center and baseline titre - pooled variance), LL = lower limit, UL = upper limit

Age\_cat is 1 for subject within age interval of 18-32 years and 2 for 33-45 years

208068 (RSV-MAT-001) Statistical Analysis Plan Final

# Template 49 Exploratory comparisons (<GMT, GMC> ratios) between RSV groups and placebo with corresponding 95% confidence interval for <RSV A neutralizing antibody titre, RSV F IgG antibody concentration> at Day 31 <PPS for immunogenicity at Day 31>

| | | | | | | | GMT ratio | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | Adjusted<br>95% CI | | Adjusted p-value |
| Antibody | Timepoint | Group description | N | <gmt,<br>GMC&gt;</gmt,<br> | Group description | <gmt,<br>GMC&gt;</gmt,<br> | Ratio order | Value | LL | UL | |
| <rsv-a nab,<br="">RSV IgG<br/>antibody&gt;</rsv-a> | PI(D8) | RSV MAT<br>120 | | | Placebo | | RSV MAT<br>120/Placebo | | | | |
| · | | RSV MAT<br>60 | | | Placebo | | RSV MAT<br>60/ Placebo | | | | |
| | | RSV MAT<br>30 | | | Placebo | | RSV MAT<br>30/Placebo | | | | |

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

Adjusted GMT = geometric mean antibody titre adjusted for age\_cat, center and baseline titre

N = Number of subjects with both pre- and post-vaccination results available

95% CI = 95% confidence interval for the GMT/GMC ratio (ANCOVA model: adjustment for age\_cat, center and

baseline titre - pooled variance), LL = lower limit, UL = upper limit

P-values were adjusted according to Dunnett for multiple comparisons to placebo

Age\_cat is 1 for subject within age interval of 18-32 years and 2 for 33-45 years

PI(D31) = Post-vaccination at Day 31

208068 (RSV-MAT-001) Statistical Analysis Plan Final

## Template 50 Descriptive statistics of <anti-RSV A neutralizing antibody titre, anti-RSV F IgG antibody concentration>at pre-vaccination, Day <8, 31, 61, 91><PPS for immunogenicity>

| | | Each Group<br>N= | | |
|---------|-------------|------------------|----|----|
| | | 95% CI | | |
| Visit | Parameters | Value | LL | UL |
| PRE | N with data | | | |
| | Mean | | | |
| | SD | | | |
| | Q1 | | | |
| | Median | | | |
| | Q3 | | | |
| PI(D8) | | | | |
| PI(D31) | | | | |
| PI(D61) | | | | |
| PI(D91) | | | | |

<each group>:

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

N = total number of subjects

N with data = number of subjects with available results

Value = value of the considered parameter

SD = standard deviation

Q1 and Q3 = 1st and 3rd quantiles

LL, UL = Exact 95% Lower and Upper confidence limits

PRE = Pre-vaccination at screening

PI(D8) = Post-vaccination at Day 8

PI(D31) = Post-vaccination at Day 31

PI(D61) = Post-vaccination at Day 61

PI(D91) = Post-vaccination at Day 91

208068 (RSV-MAT-001) Statistical Analysis Plan Final

## Template 51 Descriptive statistics of area under the curve up to Day 91 for <anti-RSV A neutralizing antibody titre, anti-RSV F IgG antibody concentration> 91><PPS for immunogenicity>

| | Each Group<br>N= | | | |
|--------------|------------------|-------|--------|----|
| | | | 95% CI | |
| Timepoint | Parameters | Value | LL | UL |
| Up to Day 91 | N with data | | | |
| | Mean<br>SD<br>Q1 | | | |
| | Median | | | |
| | Q3 | | | |

<each group>:

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Placebo = Subject receiving placebo

N = total number of subjects

N with data = number of subjects with documentation of the corresponding data

Value = value of the considered parameter

SD = standard deviation

Q1 and Q3 = 1st and 3rd quantiles

LL, UL = Exact 95% Lower and Upper confidence limits

Template 52 Assessment of trend (linear or quadratic) of dose response for <<anti-RSV A neutralizing antibody titre, anti-RSV F IgG antibody concentration> between three RSV vaccine groups at Day 31 <PPS for immunogenicity at Day 31>

| Antibody | Trend Test | N | P value |
|---|---|---|---|
| <anti-rsv a<="" td=""><td>Linear</td><td></td><td></td></anti-rsv> | Linear | | |
| Neutralizing | | | |
| Antibody, RSV | | | |
| IgG antibody> | | | |
| | Quadratic | | |

#### <each group>:

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Analysed using ANCOVA fitting treatment as fixed effect and age\_cat, center and baseline titre as covariate Contrast used for evaluating linear,quadratic> trend is

Age cat is 1 for subject within age interval of 18-32 years and 2 for 33-45 years

208068 (RSV-MAT-001) Statistical Analysis Plan Final

# Template 53 Assessment of trend (linear or quadratic) of dose response using area under curve up to Day 91 for <<anti-RSV A neutralizing antibody titre, anti-RSV F IgG antibody concentration> between three RSV vaccine groups <PPS for immunogenicity>

| Antibody | Trend Test | Ν | P value |
|---|---|---|---|
| <anti-rsv a<="" td=""><td>Linear</td><td></td><td></td></anti-rsv> | Linear | | |
| Neutralizing | | | |
| Antibody, RSV | | | |
| IgG antibody> | | | |
| | Quadratic | | |

#### <each group>:

RSV MAT 30 = Subject receiving RSVPreF3 low dose

RSV MAT 60 = Subject receiving RSVPreF3 mid dose

RSV MAT 120 = Subject receiving RSVPreF3 high dose

Analysed using ANCOVA fitting treatment as fixed effect and age\_cat, center and baseline titre as covariate Age\_cat is 1 for subject within age interval of 18-32 years and 2 for 33-45 years